CLINICAL TRIAL: NCT02688387
Title: A Phase 1 Study to Demonstrate the Relative Bioavailability of Fixed Dose Combinations of Ambrisentan and Tadalafil in Healthy Subjects
Brief Title: A Phase 1 Relative Bioavailability Study of Ambrisentan and Tadalfil Fixed Dose Combination Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Covance Harrogate (Unknown); Hammersmith Medicines Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201964
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2018-07

CONDITIONS: Hypertension, Pulmonary
Keywords: Ambrisentan; Bioavailability; Tadalafil; Fixed Dose combination
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — ambrisentan; Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 (Experimental): Enrolled subjects will receive single oral dose of 4 FDCs i.e., FDC1, FDC2, FDC3 and FDC4, and reference formulations of the 2 monotherapy components taken concurrently in the fasted state. The FDC and reference formulations contains 10 mg ambrisentan and 40 mg tadalafil. Each dosing period will be separated by 7 days wash out period.
  Interventions: Drug: FDC (ambrisentan 10 mg-tadalafil 40 mg) single dose; Drug: Reference (ambrisentan 10 mg + tadalafil 40 mg given concurrently)
- Part 2 (Experimental): Enrolled subjects will receive single oral dose of 4 FDCs i.e., FDC5, FDC6, FDC7 and FDC8, and reference formulations of the 2 monotherapy components taken concurrently in the fasted state. The FDCs and reference formulations contains 10 mg ambrisentan and 40mg Tadalafil. OR Subjects will receive single dose of two FDCs from Part 1 in fed and fasted state. Each dosing period will be separated by 7 days wash out period.
  Interventions: Drug: FDC (ambrisentan 10 mg-tadalafil 40 mg) single dose; Drug: Reference (ambrisentan 10 mg + tadalafil 40 mg given concurrently)
- Part 3 (Experimental): Enrolled subjects will receive single oral dose of 2 FDCs from Part 2 in fed and fasted state. The FDCs contains 10 mg ambrisentan and 40 mg Tadalafil. Each dosing period will be separated by 7 days wash out period.
  Interventions: Drug: FDC (ambrisentan 10 mg-tadalafil 40 mg) single dose

INTERVENTIONS:
Drug: FDC (ambrisentan 10 mg-tadalafil 40 mg) single dose — The four FDCs in part 1 will have the following formulation designation: FDC1, FDC2, FDC3 and FDC4. They are film-coated tablets. The dose will be administered orally. Study treatment for Part2 and Part 3 will be amended after Part 1 study
Drug: Reference (ambrisentan 10 mg + tadalafil 40 mg given concurrently) — Ambrisentan is a film-coated tablet. Each tablet of ambrisentan contains 10 mg of ambrisentan, approximately 95 mg of lactose (as monohydrate), 0.25 mg of lecithin and 0.11 mg of Allura red AC Aluminium Lake. Tadalafil is also a film-coated tablet. Each tablet of Tadalafil contains 20 mg tadalafil and 233 mg lactose. Both the tablets will be administered orally concurrently.
  Arms: Part 1; Part 2

SUMMARY:
This study is designed to understand the relative bioavailability (proportion of the administered dose that is absorbed into the bloodstream) of several fixed dose combinations (FDCs) tablets of ambrisentan and tadalafil for further development and to provide pharmacokinetic (PK - what the body does to the drug) data to enable a pivotal bioequivalence (BE - the relationship between two preparations of the same drug in the same dosage form that have a similar bioavailability) study. Depending on formulation work, the study will allow up to 8 new FDCs to be compared with the reference of ambrisentan and tadalafil monotherapies. The study will also evaluate up to 2 of the new formulations, that may be taken in to a BE study, to be tested for any effect on pharmacokinetics of the FDC in both fed and fasted state. This is a single centre, Phase 1, single dose, randomised, open label crossover study with 3 study parts; each study part will have up to a 5 way crossover in healthy subjects. Part 1 of the study will evaluate four formulations of the FDC (ambrisentan 10 milligram [mg] + tadalafil 40 mg) and the reference of the 2 monotherapy components taken concurrently (ambrisentan 10 mg and tadalafil 40 mg) in the fasted stated. If successful formulations are identified in this part of the study, then they will be re-formulated and tested in part 2. If no successful formulations are identified in part 1 of the study, then part 2 will be utilized to look at up to 4 new FDC formulations. However, if only two formulations, or less, are evaluated in part 2 then the FDC formulations may be tested both fed and fasted to assess food effect and part 3 will not be required. If successful formulations are identified in this study part, then up to 2 of these may be tested, for food effect, in Part 3 if not already assessed in this part. Therefore, part 3 is optional and utility is dependent on the results of the previous study parts.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 60 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests, vital signs and cardiac monitoring (ECG and 24 hour Holter). A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator, in consultation with Medical Monitor if required, judges and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >= 50 Kilogram (kg) (110 pounds [lbs]) for men and >= 45 kg (99lbs) for women and body mass index (BMI) within the range 18 - 30 kg per square metre (m^2) (inclusive)
* Male or Female. Female with non-reproductive potential defined as, Pre-menopausal females with one of the following: Documented tubal ligation or Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion or Hysterectomy or Documented Bilateral Oophorectomy, Documented Postmenopausal defined as 12 months of spontaneous amenorrhea
* Capable of giving signed informed consent.

Exclusion Criteria:

* A blood pressure <100/55 millimetre of Mercury (mm Hg).
* Haemoglobin (Hb) below normal range: Hb <133 (gram per litre) g/L for males and Hb <114 g/L for females
* Alanine amino transferase (ALT) and bilirubin >1.5 x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin is <35 percentage [%]).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Corrected QT (QTc) >450 milliseconds (msec). The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), Fridericia's formula (QTcF), and/or another method, machine-read or manually over-read.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 gram (g) of alcohol: a half-pint (~240 millilitre [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Smoking more than 5 cigarettes per week and subjects must be able to abstain from smoking for a 24 hour period prior to dose and any time whilst in the clinical unit.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at Screening or within 3 months prior to first dose of study treatment.
* A positive test for human immuno-deficiency virus (HIV) antibody
* A positive pre-study drug/alcohol screen.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within previous 3 months
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2016-03-18 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- [Derived] Okour M, Puri A, Chen G, Port K, Berni A, Khindri S, Schneider I, Tenero D. A Phase I Study to Show the Relative Bioavailability and Bioequivalence of Fixed-Dose Combinations of Ambrisentan and Tadalafil in Healthy Subjects. Clin Ther. 2019 Jun;41(6):1110-1127. doi: 10.1016/j.clinthera.2019.04.007. Epub 2019 May 4. PMID 31060740

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single dose, randomized, open-label, crossover study in healthy participants. A total of 112 healthy participants were randomized and received the study treatment. The study was conducted at a single center in the United Kingdom.
Pre-assignment Details: A total of 174 participants were screened, of which 59 were screen failures and 3 participants were reserve participants. Thus 112 participants were randomized. The study, was conducted in three parts: Part 1 (5 way crossover) and Parts 2 and 3 (A and B), followed 4 way crossover design.
Groups:
- Part 1, F2/ F3/ F1/ F4/ R: The eligible participants in the Sequence (F2/ F3/ F1/ F4/ R) received a single oral dose of fixed dose combination (FDC) for GSK3380154 (ambrisentan 10 milligram [mg] + tadalafil 40 mg). Participants received single oral dose F2 (FDC 2-GSK3380154, TAB-A, Tablet Weight 840mg/4mg Sodium laurilsulfate [SLS]) during Period 1, followed by single oral dose F3 (FDC 3- GSK3380154, TAB-A, Tablet Weight 560mg/2mg SLS) during Period 2, followed by single oral dose F1(FDC1- GSK3380154, TAB-A, Tablet Weight 840mg/2mg SLS) during Period 3, followed by a single oral dose of F4 (FDC4- GSK3380154, TAB-A, Tablet Weight 560mg/4mg SLS) during Period 4, which was followed by a single oral dose of R, a Reference- single monotherapies of 10 mg ambrisentan and 20 mg of tadalafil, taken concurrently, during Period 5. Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 7-Days.
- Part 1, R/ F1/ F4/ F2/ F3: The eligible participants in the Sequence (R/ F1/ F4/ F2/ F3), received a single oral dose of FDC for GSK3380154 (ambrisentan 10 mg + tadalafil 40 mg). Participants received single oral dose of R, a Reference- single monotherapies of 10 mg ambrisentan and 20 mg of tadalafil, taken concurrently, during Period 1, followed by single oral dose of F1(FDC1- GSK3380154, TAB-A, Tablet Weight 840mg/2mg SLS) during Period 2, followed by a single oral dose of F4 (FDC4- GSK3380154, TAB-A, Tablet Weight 560mg/4mg SLS) during Period 3, followed by single oral dose F2 (FDC 2-GSK3380154, TAB-A, Tablet Weight 840mg/4mg SLS during Period 4, followed by single oral dose F3 (FDC 3- GSK3380154, TAB-A, Tablet Weight 560mg/2mg SLS) during Period 5.Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 7-Days.
- Part 1, F4/ F3/ R/ F2/ F1: The eligible participants in the Sequence (F4/ F3/ R/ F2/ F1), received a single oral dose of FDC for GSK3380154 (ambrisentan 10 mg + tadalafil 40 mg). Participants received single oral dose of F4 (FDC4- GSK3380154, TAB-A, Tablet Weight 560mg/4mg SLS) during Period 1, followed by single oral dose F3 (FDC 3- GSK3380154, TAB-A, Tablet Weight 560mg/2mg SLS) during Period 2, followed by single oral dose of R, a Reference- single monotherapies of 10 mg ambrisentan and 20 mg of tadalafil, taken concurrently, during Period 3, followed by single oral dose F2 (FDC 2-GSK3380154, TAB-A, Tablet Weight 840mg/4mg SLS, during Period 4, followed by single oral dose of F1(FDC1- GSK3380154, TAB-A, Tablet Weight 840mg/2mg SLS), during Period 5. Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 7-Days.
- Part 1, F2/ F1/ F3/ R/ F4: The eligible participants in the Sequence (F2/ F1/ F3/ R/ F4), received a single oral dose of FDC for GSK3380154 (ambrisentan 10 mg + tadalafil 40 mg). Participants received single oral dose of F2 (FDC 2-GSK3380154, TAB-A, Tablet Weight 840mg/4mg SLS, during Period 1, followed by single oral dose of F1(FDC1- GSK3380154, TAB-A, Tablet Weight 840mg/2mg SLS), during Period 2, followed by single oral dose F3 (FDC 3- GSK3380154, TAB-A, Tablet Weight 560mg/2mg SLS) during Period 3, followed by single oral dose of R, a Reference- single monotherapies of 10 mg ambrisentan and 20 mg of tadalafil, taken concurrently, during Period 4, followed by single oral dose of F4 (FDC4- GSK3380154, TAB-A, Tablet Weight 560mg/4mg SLS) during Period 5. Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 7-Days.
- Part 1, F3/ F2/ F4/ F1/ R: The eligible participants in the Sequence (F3/ F2/ F4/ F1/ R), received a single oral dose of FDC for GSK3380154 (ambrisentan 10 mg + tadalafil 40 mg). Participants received single oral dose of F3 (FDC 3- GSK3380154, TAB-A, Tablet Weight 560mg/2mg SLS), during Period 1, followed by a single oral dose of F2 (FDC 2-GSK3380154, TAB-A, Tablet Weight 840mg/4mg SLS, during Period 2, followed by single oral dose of F4 (FDC4- GSK3380154, TAB-A, Tablet Weight 560mg/4mg SLS) during Period 3, followed by single oral dose of F1(FDC1- GSK3380154, TAB-A, Tablet Weight 840mg/2mg SLS), during Period 4, followed by single oral dose of R, a Reference- single monotherapies of 10 mg ambrisentan and 20 mg of tadalafil, taken concurrently, during Period 5. Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 7-Days.
- Part 1, F1/ F2/ R/ F3/ F4: The eligible participants in the Sequence (F1/ F2/ R/ F3/ F4), received a single oral dose of FDC for GSK3380154 (ambrisentan 10 mg + tadalafil 40 mg). Participants received single oral dose of F1(FDC1- GSK3380154, TAB-A, Tablet Weight 840mg/2mg SLS) during Period 1, followed by a single oral dose of F2 (FDC 2-GSK3380154, TAB-A, Tablet Weight 840mg/4mg SLS, during Period 2, followed by single oral dose of R, a Reference- single monotherapies of 10 mg ambrisentan and 20 mg of tadalafil, taken concurrently, during Period 3, followed by a single oral dose of F3 (FDC 3- GSK3380154, TAB-A, Tablet Weight 560mg/2mg SLS), during Period 4, followed by single oral dose of F4 (FDC4- GSK3380154, TAB-A, Tablet Weight 560mg/4mg SLS)during Period 5. Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 7-Days.
- Part 1, F3/ F4/ F2/ R/ F1: The eligible participants in the Sequence (F3/ F4/ F2/ R/ F1), , received a single oral dose of FDC for GSK3380154 (ambrisentan 10 mg + tadalafil 40 mg). Participants received single oral dose of F3 (FDC 3- GSK3380154, TAB-A, Tablet Weight 560mg/2mg SLS), during Period 1, followed by single oral dose of F4 (FDC4- GSK3380154, TAB-A, Tablet Weight 560mg/4mg SLS) during Period 2, followed by a single oral dose of F2 (FDC 2-GSK3380154, TAB-A, Tablet Weight 840mg/4mg SLS, during Period 3, followed by a single oral dose of F2 (FDC 2-GSK3380154, TAB-A, Tablet Weight 840mg/4mg SLS, during Period 4, followed by received single oral dose of F1(FDC1- GSK3380154, TAB-A, Tablet Weight 840mg/2mg SLS) during Period 5. Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 7-Days.
- Part 1, F4/ R/ F3/ F1/ F2: The eligible participants in the Sequence (F4/ R/ F3/ F1/ F2), received a single oral dose of FDC for GSK3380154 (ambrisentan 10 mg + tadalafil 40 mg). Participants received single oral dose of F4 (FDC4- GSK3380154, TAB-A, Tablet Weight 560mg/4mg SLS)during Period 1, followed by a single oral dose of R, a Reference- single monotherapies of 10 mg ambrisentan and 20 mg of tadalafil, taken concurrently during Period 2,followed by a single oral dose of F3 (FDC 3- GSK3380154, TAB-A, Tablet Weight 560mg/2mg SLS), during Period 3, followed single oral dose of F1(FDC1- GSK3380154, TAB-A, Tablet Weight 840mg/2mg SLS), during Period 4, followed by a single oral dose of F2 (FDC 2-GSK3380154, TAB-A, Tablet Weight 840mg/4mg SLS, during Period 5. Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 7-Days.
- Part 1, R/ F4/ F1/ F3/ F2: The eligible participants in the Sequence (R/ F4/ F1/ F3/ F2), received a single oral dose of FDC for GSK3380154 (ambrisentan 10 mg + tadalafil 40 mg). Participants received single oral dose of R, a Reference- single monotherapies of 10 mg ambrisentan and 20 mg of tadalafil, taken concurrently during Period 1, followed by a single oral dose of F4 (FDC4- GSK3380154, TAB-A, Tablet Weight 560mg/4mg SLS) during Period 2, followed single oral dose of F1(FDC1- GSK3380154, TAB-A, Tablet Weight 840mg/2mg SLS), during Period 3, followed by a single oral dose of F3 (FDC 3- GSK3380154, TAB-A, Tablet Weight 560mg/2mg SLS), during Period 4, followed by a s ingle oral dose of F2 (FDC 2-GSK3380154, TAB-A, Tablet Weight 840mg/4mg SLS, during Period 5. Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 7-Days.
- Part 1, F1/ R/ F2/ F4/ F3: The eligible participants in the Sequence (F1/ R/ F2/ F4/ F3), received a single oral dose of FDC for GSK3380154 (ambrisentan 10 mg + tadalafil 40 mg). Participants received single oral dose of F1(FDC1- GSK3380154, TAB-A, Tablet Weight 840mg/2mg SLS),during Period 1, followed by single oral dose of R, a Reference- single monotherapies of 10 mg ambrisentan and 20 mg of tadalafil, taken concurrently during Period 2, followed by a s ingle oral dose of F2 (FDC 2-GSK3380154, TAB-A, Tablet Weight 840mg/4mg SLS, during Period 3, followed by a single oral dose of F4 (FDC4- GSK3380154, TAB-A, Tablet Weight 560mg/4mg SLS) during Period 4, followed by a single oral dose of F3 (FDC 3- GSK3380154, TAB-A, Tablet Weight 560mg/2mg SLS), during Period 5. Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 7-Days.
- Part 2, R/ FG1/ FG3/ FG2: The eligible participants in the Sequence (R/ FG1/ FG3/ FG2) were administered the 2 monotherapies ambrisentan and tadalafil concurrently, during Period 1, this was followed by single oral dose of FDC-G1 granulation size 1 (ambrisentan 10 mg + tadalafil 40 mg), with formulation selected from Part 1, during Period 2, this was followed by the single oral dose of FDC-G2 granulation size 2 (ambrisentan 10 mg + tadalafil 40 mg) from the formulation selected from Part 1 during Period 3, this was followed by single oral dose of the FDC-G3 granulation size 3 (ambrisentan 10 mg + tadalafil 40 mg) from the formulation selected from Part 1, administered during Period 4. Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 7-Days.
- Part 2, FG1/FG2/R/ FG3: The eligible participants in the Sequence (FG1/FG2/R/ FG3) were administered single oral dose of FG1 given as FDC-G1 granulation size 1 (ambrisentan 10 mg + tadalafil 40 mg), with formulation selected from Part 1, during Period 1, this was followed by the single oral dose of FG2 given as FDC-G2 granulation size 2 (ambrisentan 10 mg + tadalafil 40 mg) from the formulation selected from Part 1 during Period 2, this was followed by the 2 monotherapies R, a Reference- single monotherapies of 10 mg ambrisentan and 20 mg of tadalafil concurrently, from the formulation selected from Part 1, given during Period 3, this was followed by single oral dose of FG3 given as FDC-G3 granulation size 3 (ambrisentan 10 mg + tadalafil 40 mg) from the formulation selected from Part 1, administered during Period 4. Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 7-Days.
- Part 2, FG2/ FG3/ FG1/ R: The eligible participants in the Sequence (FG2/ FG3/ FG1/ R), were administered single oral dose of FDC-G2 granulation size 2 (ambrisentan 10 mg + tadalafil 40 mg) from the formulation selected from Part 1 during Period 1, this was followed by single oral dose of the FDC-G3 granulation size 3 (ambrisentan 10 mg + tadalafil 40 mg) from the formulation selected from Part 1, administered during Period 2, this was followed by single oral dose of FDC-G1 granulation size 1 (ambrisentan 10 mg + tadalafil 40 mg), with formulation selected from Part 1, during Period 3, this was followed by the 2 monotherapies R, a Reference- single monotherapies of 10 mg ambrisentan and 20 mg of tadalafil concurrently, from the formulation selected from Part 1, given during Period 4. Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 7-Days.
- Part 2, FG3/ R/ FG2/ FG1: The eligible participants in the Sequence (FG3/ R/ FG2/ FG1),were administered with single oral dose of the FDC-G3 granulation size 3 (ambrisentan 10 mg + tadalafil 40 mg) from the formulation selected from Part 1, administered during Period 1, this was followed by the 2 monotherapies R, a Reference- single monotherapies of 10 mg ambrisentan and 20 mg of tadalafil concurrently, from the formulation selected from Part 1, given during Period 2, this was followed by single oral dose of FDC-G2 granulation size 2 (ambrisentan 10 mg + tadalafil 40 mg) from the formulation selected from Part 1 during Period 3, this was followed by single oral dose of FDC-G1 granulation size 1 (ambrisentan 10 mg + tadalafil 40 mg), with formulation selected from Part 1, during Period 4. Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 7-Days.
- Part 3A, X2/ R2/ R1/ X1: Eligible participants received single oral dose of X2 as FDC (ambrisentan 10 mg + tadalafil 40 mg), either FG1, FG2 or FG3 (granular formulation selected from Part 2), under fasted state during Period 1, followed by single oral dose of R2 where participants had received 2 monotherapies, for ambrisentan 10 mg and tadalafil 40 mg, as single oral dose, under fasted state during Period 2, this was followed by a single oral dose of R1 where participants had received 2 monotherapies, for ambrisentan 10 mg and tadalafil 40 mg, as single oral dose, under fed state, comprising of high fat diet during Period 3, followed by a single oral dose of X1 where participants had received FDC (ambrisentan 10 mg + tadalafil 40 mg) either FG1, FG2 or FG3 (from granular formulation selected from Part 2), under fed state, which comprised of high fat diet, during Period 4. Overall treatment period was of 4-weeks. Each dose taken either under fed or fasted condition and separated by washout period of 10-Days.
- Part 3A, ,X1/ R1/ R2/ X2: Eligible participants received single oral dose of X1 where participants had received FDC (ambrisentan 10 mg + tadalafil 40 mg) either FG1, FG2 or FG3 (from granular formulation selected from Part 2), under fed state, which comprised of a high fat diet, during Period 1, followed by single oral dose of R1 where participants had received the 2 monotherapies, for ambrisentan 10 mg and tadalafil 40 mg, as single oral dose, under fed state, comprising of high fat diet during Period 2, followed by single oral dose of R2 where participants had received 2 monotherapies, for ambrisentan 10 mg and tadalafil 40 mg, as single oral dose, under fasted state during Period 3, followed by single oral dose of X2 as FDC (ambrisentan 10 mg + tadalafil 40 mg), either FG1, FG2 or FG3 (the granular formulation selected from Part 2), under fasted state during Period 4. Overall treatment period was of 4-weeks. Each dose taken either under fed or fasted condition and separated by washout period of 10-Days.
- Part 3A, R1/ X2/ X1/ R2: Eligible participants were administered single oral dose of R1 where participants had received 2 monotherapies, for ambrisentan 10 mg and tadalafil 40 mg, as single oral dose, under fed state, comprising of high fat diet during Period 1, followed by single oral dose of X2 as FDC (ambrisentan 10 mg + tadalafil 40 mg), either FG1, FG2 or FG3 (the granular formulation selected from Part 2), under fasted state during Period 2, followed by single oral dose of X1 where participants had received FDC (ambrisentan 10 mg + tadalafil 40 mg) either FG1, FG2 or FG3 (from granular formulation selected from Part 2), under fed state, comprising high fat diet, during Period 3, followed by single oral dose of R2 where participants had received the 2 monotherapies, for ambrisentan 10 mg and tadalafil 40 mg, as single oral dose, under fasted state during Period 4. Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 10-Days.
- Part 3A, ,R2/ X1/ X2/ R1: Eligible participants were administered single oral dose of R2 where participants had received 2 monotherapies, for ambrisentan 10 mg and tadalafil 40 mg, as single oral dose, under fasted state during Period 1, followed by single oral dose of X1 where participants had received FDC (ambrisentan 10 mg + tadalafil 40 mg) either FG1, FG2 or FG3 (from granular formulation selected from Part 2), under fed state, which comprised of high fat diet, during Period 2, followed by single oral dose of X2 as FDC (ambrisentan 10 mg + tadalafil 40 mg), either FG1, FG2 or FG3 (granular formulation selected from Part 2), under fasted state during Period 3, followed by single oral dose of R1 where participants had received 2 monotherapies, for ambrisentan 10 mg and tadalafil 40 mg, as single oral dose, under fed state, comprising high fat diet during Period 4. Overall treatment period was of 4-weeks. Each dose was taken under fed or fasted condition and separated by washout period of 10-Days.
- Part 3B, Y1/ R3/ R4/ Y2: The eligible participants in the Sequence (Y1/ R3/ R4/ Y2), where participants for Y1 dose were administered a single oral dose of FDC (ambrisentan 5 mg + tadalafil 40 mg), under fasted state as a single oral dose during Period 1, this was followed by a single oral dose of R3 the participants had received the 2 monotherapies, for ambrisentan 5 mg and tadalafil 40 mg during Period 2, this was followed by a single oral dose of R4, where the participants had received the 2 monotherapies, for ambrisentan 5 mg and tadalafil 20 mg, under fasted state, during Period 3, this was followed by Y2 dose where the participants received a single oral dose of received FDC (ambrisentan 5 mg + tadalafil 20 mg), under fasted state, during Period 4. Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 10-Days.
- Part 3B, R3/ Y2/ Y1/ R4: The eligible participants in the Sequence (R3/ Y2/ Y1/ R4), where the participants for R3 dose were administered a single oral dose of the 2 monotherapies, for ambrisentan 5 mg and tadalafil 40 mg, under fasted state as a single oral dose, during Period 1, this was followed by the Y2 dose, where the participants had received FDC (ambrisentan 5 mg + tadalafil 20 mg), under fasted state as a single oral dose during Period 2, this was followed by the Y1 dose where the participants were administered a single oral dose of FDC (ambrisentan 5 mg + tadalafil 40 mg), under fasted state as a single oral dose during Period 3, this was followed by a single oral dose of R4, where the participants had received the 2 monotherapies, for ambrisentan 5 mg and tadalafil 20 mg, under fasted state, during Period 4. Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 10-Days.
- Part 3B, Y2/ R4/ R3/ Y1: The eligible participants in the Sequence (Y2/ R4/ R3/ Y1), received single oral dose of Y2 where the participants had received FDC (ambrisentan 5 mg + tadalafil 20 mg), under fasted state as a single oral dose during Period 1, this was followed by a single oral dose of R4, where the participants had received the 2 monotherapies, for ambrisentan 5 mg and tadalafil 20 mg, under fasted state, during Period 2, this was followed by a single oral dose of R3 dose where participants were administered a single oral dose of the 2 monotherapies, for ambrisentan 5 mg and tadalafil 40 mg, under fasted state, during Period 3, this was followed by the Y1 dose where the participants were administered a single oral dose of FDC (ambrisentan 5 mg + tadalafil 40 mg), under fasted state as a single oral dose during Period 4. Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 10-Days.
- Part 3B, R4/ Y1/ Y2/ R3: The eligible participants in the Sequence (R4/ Y1/ Y2/ R3), received single oral dose of R4, where the participants had received the 2 monotherapies, for ambrisentan 5 mg and tadalafil 20 mg, under fasted state, during Period 1, this was followed by the Y1 dose where the participants were administered a single oral dose of FDC (ambrisentan 5 mg + tadalafil 40 mg), under fasted state as a single oral dose during Period 2, this was followed by single oral dose of Y2 where the participants had received FDC (ambrisentan 5 mg + tadalafil 20 mg), under fasted state as a single oral dose during Period 3, this was followed by a single oral dose of R3 dose where participants were administered a single oral dose of the 2 monotherapies, for ambrisentan 5 mg and tadalafil 40 mg, under fasted state, during Period 4. Overall treatment period was of 4-weeks. Each dose was taken under fasted condition and separated by a washout period of 10-Days.
Period: Part 1, Period 1 (up to 6 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 3 | 3 | 4 | 3 | 3 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1, Washout Period 1 (7 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 3 | 3 | 3 | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 2 | 3 | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol defined stop criteria reached | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1, Period 2 (up to 6 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 3 | 2 | 3 | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol defined stop criteria reached | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1, Washout Period 2 (7 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1, Period 3 (up to 6 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1, Washout Period 3 (7 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1, Period 4 (up to 6 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1, Washout Period 4 (7 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1, Period 5 (up to 6 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2, Period 1 (up to 6 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2, Washout Period 1 (10 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2, Period 2 (up to 6 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2, Washout Period 2 (10 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2, Period 3 (up to 6 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2, Washout Period 3 (10 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2, Period 4 (up to 6 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3A, Period 1 (up to 6 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 8 | 8 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3A, Washout Period 1 (10 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3A, Period 2 (up to 6 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3A, Washout Period 2 (10 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3A, Period 3 (up to 6 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3A, Washout Period 3 (10 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3A, Period 4 (up to 6 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3B, Period 1 (up to 6 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3B, Washout Period 1 (10 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3B, Period 2 (up to 6 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3B, Washout Period 2 (10 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3B, Period 3 (up to 6 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 8 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Part 3B, Washout Period 3 (10 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 7 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Study terminated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Part 3B, Period 4 (up to 6 Days)
Arm/Group | Part 1, F2/ F3/ F1/ F4/ R | Part 1, R/ F1/ F4/ F2/ F3 | Part 1, F4/ F3/ R/ F2/ F1 | Part 1, F2/ F1/ F3/ R/ F4 | Part 1, F3/ F2/ F4/ F1/ R | Part 1, F1/ F2/ R/ F3/ F4 | Part 1, F3/ F4/ F2/ R/ F1 | Part 1, F4/ R/ F3/ F1/ F2 | Part 1, R/ F4/ F1/ F3/ F2 | Part 1, F1/ R/ F2/ F4/ F3 | Part 2, R/ FG1/ FG3/ FG2 | Part 2, FG1/FG2/R/ FG3 | Part 2, FG2/ FG3/ FG1/ R | Part 2, FG3/ R/ FG2/ FG1 | Part 3A, X2/ R2/ R1/ X1 | Part 3A, ,X1/ R1/ R2/ X2 | Part 3A, R1/ X2/ X1/ R2 | Part 3A, ,R2/ X1/ X2/ R1 | Part 3B, Y1/ R3/ R4/ Y2 | Part 3B, R3/ Y2/ Y1/ R4 | Part 3B, Y2/ R4/ R3/ Y1 | Part 3B, R4/ Y1/ Y2/ R3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7 | 6 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: In Part 1, there were 5 dosing sessions of four formulations of the FDCs (ambrisentan 10 mg + tadalafil 40 mg) (F1, F2, F3, F4) and 2 monotherapy components for ambrisentan 10 mg and tadalafil 40 mg (R) which were administered concurrently . The participants received a single oral dose of formulation or the reference during each session. All the doses were taken in fasted condition. The treatment period for Part 1 was of 4-weeks, post which there was a follow-up period of 14 days (which included 7-days washout)
- Part 2: This comprised of 4 dose sessions, of 3 different granulation sizes for a single FDC (ambrisentan 10 mg +tadalafil 40 mg) compared to the reference of the 2 monotherapy components taken concurrently (ambrisentan 10 mg & tadalafil 40 mg), to evaluate the bioavailability. This part of the study provided data for 3 granulation size forms of a single FDC formulation selected from Part 1. The participants received a single oral dose during each session. All the doses were taken in fasted condition. The treatment period for Part 2 was of 4-weeks, post which a follow-up period of 14 days (which included 7-days washout). Part 2 had FG1, FG2, FG3 which are Ambrisentan and Tadalafil FDCs (10mg/40mg). R is ambrisentan and tadalafil monotherapies taken concurrently (10mg/40mg).
- Part 3A: This comprised of 4 dose sessions of the FDC against the reference ambrisentan 10 mg + tadalafil 40mg monotherapies in the fed and fasted state, taken to evaluate the bioequivalence. The participants received a single oral dose during each session, taken under fed and fasted conditions. The fed arms of this part of the study received a standard high fat breakfast. The treatment period of Part 3A was of 4-weeks, post which a follow-up period of 14 days (which included 10-days washout). In Part 3A, X1, X2 are ambrisentan and tadalafil FDCs (10mg/40mg),where X1 is under fed state and X2 is under fasted state. R1, R2 are Ambrisentan and Tadalafil monotherapies taken concurrently(10mg/40mg), where R1 is under fed state and R2 is under fasted state.
- Part 3B: This study part comprised of 4 dose sessions which assessed the bioequivalence of the two FDC dose strengths, (ambrisentan 5 mg + tadalafil 40mg and ambrisentan 5 mg + tadalafil 20mg) against the reference ambrisentan 5 mg + tadalafil 40mg monotherapies and ambrisentan 5 mg + tadalafil 20mg monotherapies in the fasted state. The treatment period of Part 3B was of 4-weeks, post which there was a follow-up period of 14 days (which included 10-days washout). In the Part 3B, Y1, Y2 are ambrisentan and tadalafil FDCs, under fasted state, where Y1 is 5mg/40mg and Y2 is 5mg/20mg and R3, R4 are ambrisentan and tadalafil monotherapies taken concurrently, under fasted state, where R3 is 5mg/40mg and R4 is 5mg/20mg.
- Total: Total of all reporting groups
Arm/Group | Part 1 | Part 2 | Part 3A | Part 3B | Total
Number analyzed (Participants) | 26 | 21 | 33 | 32 | 112
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.7 (11.68) | 36.8 (12.07) | 37.3 (10.36) | 30.9 (12.05) | 35.5 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 1
  Male | 26 | 21 | 33 | 31 | 111
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race, Customized: Asian-Central/South Asian Heritage | 0 | 0 | 2 | 0 | 2
  Race, Customized: Asian- South East Asian heritage | 0 | 0 | 1 | 0 | 1
  Race, Customized: Black Or African American | 3 | 1 | 5 | 8 | 17
  Race, Customized: White - Arabic/North African Heritage | 0 | 0 | 0 | 1 | 1
  Race, Customized: White/Caucasian/European Heritage | 23 | 20 | 25 | 22 | 90
  Race, Customized: Multiple-Asian and White | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of Ambrisentan and Tadalafil in FDC (Ambrisentan 10 mg + Tadalafil 40 mg) and Montherapies (Ambrisentan 10 mg & Tadalafil 40 mg) - Part 1
Description: Cmax is defined as the maximum (or peak) plasma concentration that the drug achieves, after the drug has been administered. Blood samples were collected at the indicated time points for analysis of ambrisentan and tadafil. The analysis was done under fasting condition post single dose. There is no formal hypotheses tested for Part 1 of the study. The analysis was performed on Pharmacokinetic (PK) parameter population, which included all participants who provided PK parameter data.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- Part 1,Treatment F1: In the F1 arm of Part 1, the participants had received the FDC with dose session as (ambrisentan 10 mg + tadalafil 40 mg): FDC1- GSK3380154, TAB-A, Tablet Weight 840mg/2mg SLS, with reference to the 2 monotherapy components for ambrisentan 10 mg and tadalafil 40 mg, which were taken concurrently which evaluated bioavailability. This was received as a single oral dose, under fasting condition and was followed by a wash-out period of 7-days, before the start of next dose F2.
- Part 1,Treatment F2: In the F2 arm of Part 1, the participants had received the FDC with dose session as (ambrisentan 10 mg + tadalafil 40 mg): FDC2- GSK3380154, TAB-A, Tablet Weight 840mg/4mg SLS, with reference to the 2 monotherapy components for ambrisentan 10 mg and tadalafil 40 mg, which were taken concurrently which evaluated bioavailability. This was received as a single oral dose, under fasting condition and was followed by a wash-out period of 7-days, before the start of next dose F3.
- Part 1,Treatment F3: In the F3 arm of Part 1, the participants had received the FDC with dose session as (ambrisentan 10 mg + tadalafil 40 mg): GSK3380154, TABA, Tablet Weight 560mg/2mg SLS, with reference to the 2 monotherapy components for ambrisentan 10 mg and tadalafil 40 mg, which were taken concurrently, which evaluated bioavailability. This was received as a single oral dose, under fasting condition and was followed by a wash-out period of 7-days, before the start of next dose F4.
- Part 1,Treatment F4: In the F4 arm of Part 1, the participants had received the FDC with dose session as (ambrisentan 10 mg + tadalafil 40 mg): GSK3380154, TAB-A, Tablet Weight 560mg/4mg SLS, with reference to the 2 monotherapy components for ambrisentan 10 mg and tadalafil 40 mg, which were taken concurrently, which evaluated bioavailability. This was received as a single oral dose, under fasting condition and was followed by a wash-out period of 7-days, before the start of next dose R.
- Part 1, Treatment R: In the R arm of Part 1, the participants had received the 2 monotherapies ambrisentan 10 mg and tadalafil 40 mg concurrently. The tablets were taken as single oral dose, under fasting condition and was followed by a wash-out period of 7-days.
Arm/Group | Part 1,Treatment F1 | Part 1,Treatment F2 | Part 1,Treatment F3 | Part 1,Treatment F4 | Part 1, Treatment R
Number analyzed (Participants) | 21 | 23 | 23 | 22 | 21
Nanogram per milliliter
  Ambrisentan, Cmax | 766.29 (18.2) | 685.33 (20.5) | 738.49 (22.1) | 722.57 (27.7) | 755.37 (28.9)
  Tadalafil, Cmax | 581.41 (27.6) | 595.47 (22.3) | 588.11 (24.5) | 590.36 (21.4) | 567.62 (18.0)

2. Primary Outcome: Area Under the Plasma Concentration Time Curve (AUC) From Time Zero to Infinite (Inf) Time, AUC (0-inf) of Ambrisentan and Tadalafil in FDC (Ambrisentan 10 mg + Tadalafil 40 mg) and Montherapies (Ambrisentan 10 mg & Tadalafil 40 mg) - Part 1
Description: AUC (0- inf), is defined as area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity for ambrisentan and tadafil. Blood samples were collected at the indicated time-points. The analysis was done under fasting condition post single dose. There is no formal hypothesis tested for Part 1 of the study.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 1,Treatment F1 | Part 1,Treatment F2 | Part 1,Treatment F3 | Part 1,Treatment F4 | Part 1, Treatment R
Number analyzed (Participants) | 21 | 23 | 23 | 22 | 21
Hour*nanogram per milliliter
  Ambrisentan, (AUC 0 - inf) | 5566.06 (23.8) | 5556.44 (25.9) | 5788.91 (25.8) | 6007.57 (23.7) | 5746.73 (20.8)
  Tadalafil, (AUC 0 - inf) | 13408.30 (41.3) | 14415.47 (41.8) | 14545.28 (38.4) | 14418.35 (37.8) | 13955.85 (36.2)

3. Primary Outcome: AUC From Time of Dose to Last Measurable Concentration (AUC [0-t]), in FDC, (Ambrisentan 10 mg + Tadalafil 40 mg) Relative to Reference Monotherapies Tested (Ambrisentan 10 mg & Tadalafil 40 mg), Under Fasting- Part 1
Description: AUC (0-t), was defined as, the AUC measured from the time of dose to the last measurable concentration. Blood samples of 2.7 mL and 2 mL, were collected for ambrisentan and tadafil respectively. The plasma samples at Part 1, were collected at the time-points pre-dose, 0.5 hours, 1, 1.5, 2, 2.5, 4, 8, 12, 24, 36, 48 and 72 hours. The analysis was done under fasting condition post single dose. The PK Parameter Population was used for analysis. There is no formal hypotheses tested for Part 1 of the study.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 1,Treatment F1 | Part 1,Treatment F2 | Part 1,Treatment F3 | Part 1,Treatment F4 | Part 1, Treatment R
Number analyzed (Participants) | 21 | 23 | 23 | 22 | 21
Hour*nanogram per milliliter
  Ambrisentan, (AUC 0- t) | 5418.03 (22.9) | 5434.88 (25.3) | 5655.75 (25.5) | 5858.18 (22.9) | 5605.58 (20.2)
  Tadalafil, (AUC 0- t) | 12469.86 (37.1) | 13307.95 (37.4) | 13376.86 (34.8) | 13238.89 (33.4) | 12805.01 (32.2)

4. Primary Outcome: Cmax of Ambrisentan and Tadalafil in FDC (Ambrisentan 10 mg + Tadalafil 40 mg) and Montherapies (Ambrisentan 10 mg & Tadalafil 40 mg) - Part 2
Description: Cmax is defined as the maximum (or peak) plasma concentration that the drug achieves, after the drug has been administered. Blood samples were collected at the indicated time-points, of Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose. The analysis was done under fasting condition post single dose. There is no formal hypotheses tested for Part 2 of the study. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- Part 2, Treatment R: Participants were administered 2 monotherapies, ambrisentan and tadalafil concurrently. The tablets were taken as single oral dose, under fasting condition and was followed by a wash-out period of 7-days.
- Part 2, Treatment FG1: Participants were administered the FDC-G1 granulation size 1 (ambrisentan 10 mg + tadalafil 40 mg) , from the formulation selected from Part 1. FG1 was administered as a single oral dose, under fasting condition and was followed by a wash-out period of 7-days, before the start of next dose FG2.
- Part 2, Treatment FG2: Participants were administered the FDC-G2 granulation size 2 (ambrisentan 10 mg + tadalafil 40 mg) from the formulation selected from Part 1. FG2 was administered as a single oral dose, under fasting condition and was followed by a wash-out period of 7-days, before the start of next dose FG3.
- Part 2, Treatment FG3: Participants were administered the FDC-G3 granulation size 3 (ambrisentan 10 mg + tadalafil 40 mg) from the formulation selected from Part 1. FG3 was received as a single oral dose, under fasting condition and was followed by a wash-out period of 7-days, before the start of next dose R.
Arm/Group | Part 2, Treatment R | Part 2, Treatment FG1 | Part 2, Treatment FG2 | Part 2, Treatment FG3
Number analyzed (Participants) | 21 | 20 | 20 | 20
Nanogram per milliliter
  Ambrisentan, (n=21,20,20,20) | 710.90 (28.2) | 720.79 (21.1) | 748.63 (22.9) | 726.15 (31.4)
  Tadalafil, (n=20,20,20,20): number analyzed (Participants) | 20 | 20 | 20 | 20
  Tadalafil, (n=20,20,20,20) | 537.80 (27.6) | 561.60 (28.4) | 550.78 (28.6) | 553.31 (20.5)

5. Primary Outcome: AUC (0 - Inf) for FDC, (Ambrisentan 10 mg + Tadalafil 40 mg) Relative to Reference Monotherapies Tested (Ambrisentan 10 mg & Tadalafil 40 mg), Under Fasting- Part 2
Description: AUC (0- inf), is defined as area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity for ambrisentan and tadafil. Blood samples of 2.7 mL and 2 mL were collected for ambrisentan and tadafil respectively. The plasma samples for Part 2, were collected at the time-points pre-dose, 0.5 hours, 1, 1.5, 2, 2.5, 4, 8, 12, 24, 36, 48 and 72 hours post-dose. The analysis, was done under fasting condition post single dose. PK parameter Populatio was used for analysis. There is no formal hypotheses tested for Part 2 of the study. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 2, Treatment R | Part 2, Treatment FG1 | Part 2, Treatment FG2 | Part 2, Treatment FG3
Number analyzed (Participants) | 21 | 20 | 20 | 20
Hour*nanogram per milliliter
  Ambrisentan, AUC (0-inf) (n=21,20,20,20) | 6029.19 (29.6) | 6179.41 (27.2) | 6189.22 (29.5) | 6201.40 (25.7)
  Tadalafil, AUC ( 0 - inf) (n=20,20,20,20): number analyzed (Participants) | 20 | 20 | 20 | 20
  Tadalafil, AUC ( 0 - inf) (n=20,20,20,20) | 14006.59 (46.7) | 14443.86 (44.8) | 14502.37 (40.5) | 14457.33 (40.5)

6. Primary Outcome: AUC (0-t) for FDC, (Ambrisentan 10 mg + Tadalafil 40 mg) Relative to Reference Monotherapies Tested (Ambrisentan 10 mg & Tadalafil 40 mg), Under Fasting- Part 2
Description: AUC (0-t), was defined as, the AUC measured from the time of dose to the last measurable concentration. Blood samples of 2.7 mL and 2 mL, were collected for ambrisentan and tadafil respectively. The plasma samples for Part 2, were collected at the time-points pre-dose, 0.5 hours, 1, 1.5, 2, 2.5, 4, 8, 12, 24, 36, 48 and 72 hours. The analysis was done under fasting condition post single dose. PK parameter Population was used for analysis. There is no formal hypotheses tested for Part 2 of the study. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 2, Treatment R | Part 2, Treatment FG1 | Part 2, Treatment FG2 | Part 2, Treatment FG3
Number analyzed (Participants) | 21 | 20 | 20 | 20
Hour*nanogram per milliliter
  Ambrisentan, (n=21,20,20,20) | 5893.74 (29.4) | 6016.62 (27.1) | 6051.83 (29.6) | 6015.11 (25.9)
  Tadalafil, (n=20,20,20,20): number analyzed (Participants) | 20 | 20 | 20 | 20
  Tadalafil, (n=20,20,20,20) | 12832.91 (39.6) | 13149.19 (37.5) | 13305.50 (35.2) | 13275.08 (33.3)

7. Primary Outcome: Cmax for Ambrisentan and Tadalafil, Following Candidate FDC (Ambrisentan 10 mg + Tadalafil 40 mg) Relative to Reference Monotherapies Tested (Ambrisentan 10 mg & Tadalafil 40 mg), Under Fed and Fasted Conditions-Part 3A
Description: Cmax is defined as the maximum (or peak) plasma concentration that the drug achieves, after the drug has been administered. Blood samples of 2.7 mL and 2 mL were collected for ambrisentan and tadafil respectively. The plasma samples for Part 3A, were collected at the time-points pre-dose, 0.5 hours, 1, 1.5, 2, 2.5, 4, 8, 12, 24, 36, 48 and 72 hours post-dose. The analysis was done under fed and fasting condition post single dose. PK parameter population was used.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- Part 3A,Treatment X1: In the X1 arm of Part 3A, which evaluated the bioequivalence, the participants had received FDC (ambrisentan 10 mg + tadalafil 40 mg) either FG1, FG2 or FG3 (from granular formulation selected from Part 2), under fed state as a single oral dose. The fed state, participants received a high fat diet. This was followed by a wash-out period of 10-days, before the start of next dose X2.
- Part 3A,Treatment X2: In the X2 arm of Part 3A, which evaluated the bioequivalence, the participants had received FDC (ambrisentan 10 mg + tadalafil 40 mg), either FG1, FG2 or FG3 (the granular formulation selected from Part 2), under fasted state as a single oral dose. This was followed by a wash-out period of 10-days, before the start of next dose R1.
- Part 3A,Treatment R1: In the R1 arm, of Part 3A, the participants had received the 2 monotherapies, for ambrisentan 10 mg and tadalafil 40 mg, as single oral dose, under fed state. Fed state comprised of high fat diet. This was followed by a wash-out period of 10-days, before the start of next dose R2.
- Part 3A,Treatment R2: In the R2 arm, of Part 3A, the participants had received the 2 monotherapies, for ambrisentan 10 mg and tadalafil 40 mg, as single oral dose, under fasted state. This was followed by a wash-out period of 10-days.
Arm/Group | Part 3A,Treatment X1 | Part 3A,Treatment X2 | Part 3A,Treatment R1 | Part 3A,Treatment R2
Number analyzed (Participants) | 32 | 33 | 32 | 32
Nanogram per milliliter
  Ambrisentan, Cmax | 550.02 (30.9) | 756.60 (24.1) | 515.61 (33.4) | 728.32 (29.8)
  Tadalafil, Cmax | 525.10 (26.5) | 508.72 (24.9) | 533.67 (19.5) | 520.62 (21.1)
Statistical Analysis 1: Comparison: Part 3A,Treatment X1 vs Part 3A,Treatment R1; Test type: Equivalence — Part 3A of the study is designed to test the bioequivalence of a FDC of ambrisentan 10 mg + tadalafil 40 mg (test) relative to reference monotherapies of ambrisentan 10 mg & tadalafil 40 mg taken concurrently (reference) in healthy participants in both the fed and fasted states; Ratio = 1.0667, 90% CI 2-sided [0.9657 to 1.1784] — X1 Vs R1, ambrisentan
Statistical Analysis 2: Comparison: Part 3A,Treatment X2 vs Part 3A,Treatment R2; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; Ratio = 1.0353, 90% CI 2-sided [0.9293 to 1.1534] — X2 Vs R2, ambrisentan
Statistical Analysis 3: Comparison: Part 3A,Treatment X1 vs Part 3A,Treatment R1; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; Ratio = 0.9839, 90% CI 2-sided [0.9288 to 1.0423] — X1 Vs R1, tadalafil
Statistical Analysis 4: Comparison: Part 3A,Treatment X2 vs Part 3A,Treatment R2; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; Ratio = 0.9656, 90% CI 2-sided [0.9151 to 1.0188] — X2 Vs R2, tadalafil

8. Primary Outcome: AUC (0-inf) for Ambrisentan and Tadalafil, Following Candidate FDC (Ambrisentan 10 mg + Tadalafil 40 mg) Relative to Reference Monotherapies Tested (Ambrisentan 10 mg & Tadalafil 40 mg), Under Fed and Fasted Conditions-3A
Description: AUC (0- inf), is defined as area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity for ambrisentan and tadafil. Blood samples of 2.7 mL and 2 mL were collected for ambrisentan and tadafil respectively. The plasma samples for Part 3A, were collected at the time-points pre-dose, 0.5 hours, 1, 1.5, 2, 2.5, 4, 8, 12, 24, 48 and 72 hours post-dose. The analysis, was done under fed and fasting conditions post single dose. PK parameter population was used.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 3A,Treatment X1 | Part 3A,Treatment X2 | Part 3A,Treatment R1 | Part 3A,Treatment R2
Number analyzed (Participants) | 32 | 33 | 32 | 32
Hour*nanogram per milliliter
  Ambrisentan, AUC (0-inf) | 6075.51 (26.1) | 6231.48 (25.1) | 5898.72 (27.7) | 6155.60 (24.4)
  Tadalafil, AUC (0-inf) | 16086.66 (41.5) | 14856.32 (40.0) | 16596.18 (37.8) | 14612.84 (41.5)
Statistical Analysis 1: Comparison: Part 3A,Treatment X1 vs Part 3A,Treatment R1; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; Ratio = 1.0300, 90% CI 2-sided [0.9965 to 1.0646] — X1 Vs R1, ambrisentan
Statistical Analysis 2: Comparison: Part 3A,Treatment X2 vs Part 3A,Treatment R2; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; Ratio = 1.0141, 90% CI 2-sided [0.9820 to 1.0473] — X2 Vs R2, ambrisentan
Statistical Analysis 3: Comparison: Part 3A,Treatment X1 vs Part 3A,Treatment R1; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; Ratio = 0.9693, 90% CI 2-sided [0.9310 to 1.0092] — X1 Vs R1, tadalafil
Statistical Analysis 4: Comparison: Part 3A,Treatment X2 vs Part 3A,Treatment R2; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; Ratio = 1.0157, 90% CI 2-sided [0.9553 to 1.0799] — X2 Vs R2, tadalafil

9. Primary Outcome: AUC (0-t) for Ambrisentan and Tadalafil, Following Candidate FDC (Ambrisentan 10 mg + Tadalafil 40 mg) Relative to Reference Monotherapies Tested (Ambrisentan 10 mg & Tadalafil 40 mg), Under Fed and Fasted Conditions-Part 3A
Description: AUC (0-t), was defined as, the AUC measured from the time of dose to the last measurable concentration. Blood samples of 2.7 mL and 2 mL, were collected for ambrisentan and tadafil respectively. The plasma samples for Part 3A, were collected at the time-points pre-dose, 0.5 hours, 1, 1.5, 2, 2.5, 4, 8, 12, 24, 36, 48 and 72 hours post-dose. The analysis was done under fed and fasting condition post single dose. PK parameter population was used.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 3A,Treatment X1 | Part 3A,Treatment X2 | Part 3A,Treatment R1 | Part 3A,Treatment R2
Number analyzed (Participants) | 32 | 33 | 32 | 32
Hour*nanogram per milliliter
  Ambrisentan, AUC (0-t) | 5926.87 (25.7) | 6090.74 (24.8) | 5766.71 (27.4) | 6012.51 (24.0)
  Tadalafil, AUC (0-t) | 14366.73 (33.7) | 13320.79 (32.4) | 14946.32 (31.1) | 13114.00 (32.6)
Statistical Analysis 1: Comparison: Part 3A,Treatment X1 vs Part 3A,Treatment R1; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; Ratio = 1.0278, 90% CI 2-sided [0.9943 to 1.0623] — X1 Vs R1, ambrisentan
Statistical Analysis 2: Comparison: Part 3A,Treatment X2 vs Part 3A,Treatment R2; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; Ratio = 1.0144, 90% CI 2-sided [0.9832 to 1.0466] — X2 Vs R2, ambrisentan
Statistical Analysis 3: Comparison: Part 3A,Treatment X1 vs Part 3A,Treatment R1; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; Ratio = 0.9612, 90% CI 2-sided [0.9265 to 0.9972] — X1 Vs R1, tadalafil
Statistical Analysis 4: Comparison: Part 3A,Treatment X2 vs Part 3A,Treatment R2; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; Ratio = 1.0122, 90% CI 2-sided [0.9562 to 1.0715] — X2 Vs R2, tadalafil

10. Primary Outcome: Cmax for Ambrisentan and Tadalafil, FDCs (Ambrisentan 5 mg + Tadalafil 40 mg) Relative to Reference Monotherapies Tested (Ambrisentan 5 mg & Tadalafil 40 mg) Under Fasted Conditions-3B
Description: Cmax is defined as the maximum (or peak) plasma concentration that the drug achieves, after the drug has been administered. Blood samples of 2.7 mL and 2 mL were collected for ambrisentan and tadafil respectively. The plasma samples for Part 3B, were collected at the time-points pre-dose, 0.5 hours, 1, 1.5, 2, 2.5, 4, 8, 12, 24, 36, 48 and 72 hours post-dose. The analysis was done under fasting condition post single dose.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- Part 3B,Treatment Y1: In the Y1 arm of Part 3B, which evaluated bioequivalence, the participants had received FDC (ambrisentan 5 mg + tadalafil 40 mg), under fasted state as a single oral dose. This was followed by a wash-out period of 10-days, before the start of next dose Y2
- Part 3B,Treatment R3: In the R3 arm of Part 3B, which evaluated bioequivalence, the participants had received the 2 monotherapies, for ambrisentan 5 mg and tadalafil 40 mg, under fasted state as a single oral dose. This was followed by a wash-out period of 10-days, before the start of next dose of R4.
Arm/Group | Part 3B,Treatment Y1 | Part 3B,Treatment R3
Number analyzed (Participants) | 30 | 31
Nanogram per milliliter
  Ambrisentan, Cmax | 375.87 (23.0) | 380.47 (26.2)
  Tadalafil, Cmax | 488.36 (19.7) | 511.80 (28.3)
Statistical Analysis 1: Comparison: Part 3B,Treatment Y1 vs Part 3B,Treatment R3; Test type: Equivalence — Part 3B of the study is set to establish bioequivalence between the Fixed Dose Combination of an additional two dose strengths (ambrisentan 5 mg + tadalafil 40 mg and ambrisentan 5 mg + tadalafil 20 mg); Ratio = 1.0153, 90% CI 2-sided [0.9348 to 1.1027] — Y1 Vs R3, ambrisentan
Statistical Analysis 2: Comparison: Part 3B,Treatment Y1 vs Part 3B,Treatment R3; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; Ratio = 0.9758, 90% CI 2-sided [0.9044 to 1.0529] — Y1 Vs R3, tadalafil

11. Primary Outcome: AUC (0-inf) for Ambrisentan and Tadalafil, FDCs (Ambrisentan 5 mg + Tadalafil 40 mg) Relative to Reference Monotherapies Tested (Ambrisentan 5 mg & Tadalafil 40 mg) Under Fasted Conditions-3B
Description: AUC (0- inf), is defined as area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity for ambrisentan and tadafil. Blood samples of 2.7 mL and 2 mL were collected for ambrisentan and tadafil respectively. The plasma samples for Part 3B, were collected at the time-points pre-dose, 0.5 hours, 1, 1.5, 2, 2.5, 4, 8, 12, 24, 36,48 and 72 hours post-dose. The analysis was done under fasting condition post single dose. PK Parameter Population was used for analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour nanogram per milliliter
Arm/Group | Part 3B,Treatment Y1 | Part 3B,Treatment R3
Number analyzed (Participants) | 30 | 31
Hour nanogram per milliliter
  Ambrisentan AUC (0-inf) | 3397.51 (19.7) | 3277.81 (20.8)
  Tadalafil, AUC (0-inf) | 14724.34 (39.7) | 14938.29 (40.7)
Statistical Analysis 1: Comparison: Part 3B,Treatment Y1 vs Part 3B,Treatment R3; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; Ratio = 1.0390, 90% CI 2-sided [1.0168 to 1.0617] — Y1 Vs R3, ambrisentan
Statistical Analysis 2: Comparison: Part 3B,Treatment Y1 vs Part 3B,Treatment R3; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; Ratio = 0.9806, 90% CI 2-sided [0.9106 to 1.0560] — Y1 Vs R3, tadalafil

12. Primary Outcome: AUC (0-t) for Ambrisentan and Tadalafil, FDCs (Ambrisentan 5 mg + Tadalafil 40 mg) Relative to Reference Monotherapies Tested (Ambrisentan 5 mg & Tadalafil 40 mg) Under Fasted Conditions-3B
Description: AUC (0-t), was defined as, the AUC measured from the time of dose to the last measurable concentration. Blood samples of 2.7 mL and 2 mL, were collected for ambrisentan and tadafil respectively. The plasma samples for Part 3B, were collected at the time-points pre-dose, 0.5 hours, 1, 1.5, 2, 2.5, 4, 8, 12, 24, 36, 48 and 72 hours post-dose. The analysis was done under fasting condition post single dose. PK parameter population was used for analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 3B,Treatment Y1 | Part 3B,Treatment R3
Number analyzed (Participants) | 30 | 31
Hour*nanogram per milliliter
  Ambrisentan, AUC (0-t) | 3297.16 (19.8) | 3190.51 (20.3)
  Tadalafil, AUC (0-t) | 13119.89 (31.0) | 13325.63 (35.0)
Statistical Analysis 1: Comparison: Part 3B,Treatment Y1 vs Part 3B,Treatment R3; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; Ratio = 1.0365, 90% CI 2-sided [1.0138 to 1.0596] — Y1 Vs R3, ambrisentan
Statistical Analysis 2: Comparison: Part 3B,Treatment Y1 vs Part 3B,Treatment R3; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; Ratio = 0.9821, 90% CI 2-sided [0.9145 to 1.0547] — Y1 Vs R3, tadalafil

13. Primary Outcome: Cmax for Ambrisentan and Tadalafil, FDCs (Ambrisentan 5 mg + Tadalafil 20 mg) Relative to Reference Monotherapies Tested (Ambrisentan 5 mg & Tadalafil 20 mg) Under Fasted Conditions-3B
Description: Cmax is defined as the maximum (or peak) plasma concentration that the drug achieves, after the drug has been administered. Blood samples of 2.7 mL and 2 mL were collected for ambrisentan and tadafil respectively. The plasma samples for Part 3B, were collected at the time-points pre-dose, 0.5 hours, 1, 1.5, 2, 2.5, 4, 8, 12, 24, 36, 48 and 72 hours post-dose. The analysis was done under fasting condition post single dose. PK parameter population was used.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- Part 3B,Treatment Y2: In the Y2 arm of Part 3B, which evaluated bioequivalence, the participants had received FDC (ambrisentan 5 mg + tadalafil 20 mg), under fasted state as a single oral dose. This was followed by a wash-out period of 10-days, before the start of next dose R3.
- Part 3B,Treatment R4: In the R4 arm of Part 3B, which evaluated bioequivalence, the participants had received the 2 monotherapies, for ambrisentan 5 mg and tadalafil 20 mg, under fasted state as a single oral dose. This was followed by a wash-out period of 10-days.
Arm/Group | Part 3B,Treatment Y2 | Part 3B,Treatment R4
Number analyzed (Participants) | 31 | 30
Nanogram per milliliter
  Ambrisentan, Cmax | 405.89 (25.1) | 358.89 (24.5)
  Tadalafil, Cmax | 340.63 (23.1) | 303.74 (22.5)
Statistical Analysis 1: Comparison: Part 3B,Treatment Y2 vs Part 3B,Treatment R4; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; Ratio = 1.1176, 90% CI 2-sided [1.0166 to 1.2287] — Y2 Vs R4, ambrisentan
Statistical Analysis 2: Comparison: Part 3B,Treatment Y2 vs Part 3B,Treatment R4; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; Ratio = 1.1196, 90% CI 2-sided [1.0429 to 1.2019] — Y2 Vs R4, tadalafil

14. Primary Outcome: AUC (0-inf) for Ambrisentan and Tadalafil, FDCs (Ambrisentan 5 mg + Tadalafil 20 mg) Relative to Reference Monotherapies Tested (Ambrisentan 5 mg & Tadalafil 20 mg) Under Fasted Conditions-3B
Description: AUC (0- inf), is defined as area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity for ambrisentan and tadafil. Blood samples of 2.7 mL and 2 mL were collected for ambrisentan and tadafil respectively. The plasma samples for Part 3B, were collected at the time-points pre-dose, 0.5 hours, 1, 1.5, 2, 2.5, 4, 8, 12, 24, 36, 48 and 72 hours post-dose. The analysis, was done under fasting conditions post single dose. PK parameter population was used for analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 3B,Treatment Y2 | Part 3B,Treatment R4
Number analyzed (Participants) | 31 | 30
Hour*nanogram per milliliter
  Ambrisentan AUC (0-inf) | 3347.76 (20.9) | 3205.51 (20.6)
  Tadalafil, AUC (0-inf) | 7962.14 (32.2) | 7748.47 (32.6)
Statistical Analysis 1: Comparison: Part 3B,Treatment Y2 vs Part 3B,Treatment R4; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; Ratio = 1.0353, 90% CI 2-sided [1.0009 to 1.0710] — Y2 Vs R4, ambrisentan
Statistical Analysis 2: Comparison: Part 3B,Treatment Y2 vs Part 3B,Treatment R4; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; Ratio = 1.0362, 90% CI 2-sided [0.9910 to 1.0834] — Y2 Vs R4, tadalafil

15. Primary Outcome: AUC (0-t) for Ambrisentan and Tadalafil, FDCs (Ambrisentan 5 mg + Tadalafil 20 mg) Relative to Reference Monotherapies Tested (Ambrisentan 5 mg & Tadalafil 20 mg) Under Fasted Conditions- Part 3B
Description: as for outcome 12
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 3B,Treatment Y2 | Part 3B,Treatment R4
Number analyzed (Participants) | 31 | 30
Hour*nanogram per milliliter
  Ambrisentan AUC (0-t) | 3254.70 (21.0) | 3116.10 (20.3)
  Tadalafil, AUC (0-t) | 7264.28 (26.6) | 7076.48 (27.4)
Statistical Analysis 1: Comparison: Part 3B,Treatment Y2 vs Part 3B,Treatment R4; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; Ratio = 1.0351, 90% CI 2-sided [1.0002 to 1.0713] — Y2 Vs R4, ambrisentan
Statistical Analysis 2: Comparison: Part 3B,Treatment Y2 vs Part 3B,Treatment R4; Test type: Equivalence — [test comment as in outcome 10, analysis 1]; Ratio = 1.0324, 90% CI 2-sided [0.9929 to 1.0734] — Y2 Vs R4, tadalafil

16. Secondary Outcome: Time Taken to Reach Maximum Concentration (Tmax) for Ambrisentan and Tadalafil in FDC and Reference Treatment - Part 1
Description: Serial blood samples were collected at the indicated time-points. In Part 3A, tmax was determined for ambrisentan and tadalafil when administered in FDC (10mg/40mg) under fed state and fasted state and as reference monotherapies (ambrisentan 10 mg and tadalafil 40 mg). PK parameter population was used to measure the tmax.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK parameter Population.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 1,Treatment F1 | Part 1,Treatment F2 | Part 1,Treatment F3 | Part 1,Treatment F4 | Part 1, Treatment R
Number analyzed (Participants) | 21 | 23 | 23 | 22 | 21
Hour
  Ambrisentan, Tmax | 1.000 [0.50 to 8.23] | 1.500 [0.53 to 4.00] | 1.500 [0.52 to 4.00] | 1.500 [0.57 to 4.05] | 1.500 [0.50 to 4.00]
  Tadafil, Tmax | 1.500 [0.50 to 8.23] | 2.000 [0.50 to 8.03] | 2.000 [0.50 to 8.00] | 2.000 [0.50 to 8.00] | 1.500 [0.50 to 4.00]

17. Secondary Outcome: Time Taken to Reach Maximum Concentration (Tmax) for Ambrisentan and Tadalafil in FDC and Reference Treatment - Part 2
Description: Serial blood samples were collected at the indicated time-points. In Part 3A, tmax was determined for ambrisentan and tadalafil when administered in FDC (10mg/40mg) under fed state and fasted state and as reference monotherapies (ambrisentan 10 mg and tadalafil 40 mg). PK parameter population was used to measure the tmax. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK parameter population.
Measure: Median (Full Range); unit: hour
Arm/Group | Part 2, Treatment R | Part 2, Treatment FG1 | Part 2, Treatment FG2 | Part 2, Treatment FG3
Number analyzed (Participants) | 21 | 20 | 20 | 20
hour
  Ambrisentan, Tmax (n=21,20,20,20) | 1.500 [0.50 to 4.03] | 1.500 [0.50 to 4.00] | 1.500 [0.50 to 4.00] | 1.508 [1.00 to 8.00]
  Tadafil, Tmax (n=20,20,20,20): number analyzed (Participants) | 20 | 20 | 20 | 20
  Tadafil, Tmax (n=20,20,20,20) | 2.017 [0.50 to 8.02] | 1.750 [0.50 to 8.08] | 2.000 [0.50 to 8.00] | 2.000 [0.50 to 12.10]

18. Secondary Outcome: Time Taken to Reach Maximum Concentration (Tmax) for Ambrisentan and Tadalafil in FDC and Reference Treatment - Part 3A
Description: as for outcome 16
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK parameter Population.
Measure: Median (Full Range); unit: Hour
Groups:
- Part 3A,Treatment R1: In the R1 arm, of Part 3A, , the participants had received the 2 monotherapies, for ambrisentan 10 mg and tadalafil 40 mg, as single oral dose, under fed state. Fed state comprised of high fat diet. This was followed by a wash-out period of 10-days, before the start of next dose R2.
Arm/Group | Part 3A,Treatment X1 | Part 3A,Treatment X2 | Part 3A,Treatment R1 | Part 3A,Treatment R2
Number analyzed (Participants) | 32 | 33 | 32 | 32
Hour
  Ambrisentan, Tmax | 4.00 [1.00 to 12.00] | 1.500 [0.50 to 4.00] | 4.00 [1.00 to 12.15] | 2.000 [1.00 to 4.00]
  Tadafil, Tmax | 8.000 [0.50 to 12.02] | 2.500 [0.50 to 12.02] | 8.000 [1.50 to 12.15] | 2.258 [0.50 to 8.03]

19. Secondary Outcome: Time Taken to Reach Maximum Concentration (Tmax) for Ambrisentan and Tadalafil in FDC and Reference Treatment - Part 3B
Description: Serial blood samples were collected at the indicated time-points. In Part 3B, tmax was determined for ambrisentan and tadalafil when administered in FDC (10mg/40mg) under fed state and fasted state and as reference monotherapies (ambrisentan 10 mg and tadalafil 40 mg). PK parameter population was used to measure the tmax.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK parameter Population.
Measure: Median (Full Range); unit: Hour
Arm/Group | Part 3B,Treatment Y1 | Part 3B,Treatment Y2 | Part 3B,Treatment R3 | Part 3B,Treatment R4
Number analyzed (Participants) | 30 | 31 | 31 | 30
Hour
  Ambrisentan, Tmax | 1.767 [1.00 to 4.03] | 1.500 [1.00 to 8.00] | 2.000 [1.00 to 8.00] | 1.758 [1.00 to 8.00]
  Tadafil, Tmax | 2.500 [0.50 to 8.00] | 1.500 [0.50 to 8.00] | 2.500 [0.50 to 8.00] | 2.008 [0.50 to 8.00]

20. Secondary Outcome: Plasma Half Life (t1/2) for Ambrisentan and Tadalafil in FDC and Reference Treatment Under Fed and Fasted Condition- Part1
Description: t1/2 is defined as the time required by the concentration of the drug to reach half of its original value.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Groups:
- Part 1,Treatment F1: In the F1 arm of Part 1, the participants had received the FDC with dose session as (ambrisentan 10 milligram (mg) + tadalafil 40 mg): FDC1- GSK3380154, TAB-A, Tablet Weight 840mg/2mg Sodium laurilsulfate (SLS), with reference to the 2 monotherapy components for ambrisentan 10 mg and tadalafil 40 mg, which were taken concurrently which evaluated bioavailability. This was received as a single oral dose, under fasting condition and was followed by a wash-out period of 7-days, before the start of next dose F2.
- Part 1,Treatment F2: In the F2 arm of Part 1, the participants had received the FDC with dose session as (ambrisentan 10 milligram (mg) + tadalafil 40 mg): FDC2- GSK3380154, TAB-A, Tablet Weight 840mg/4mg SLS, with reference to the 2 monotherapy components for ambrisentan 10 mg and tadalafil 40 mg, which were taken concurrently which evaluated bioavailability. This was received as a single oral dose, under fasting condition and was followed by a wash-out period of 7-days, before the start of next dose F3.
- Part 1,Treatment F3: In the F3 arm of Part 1, the participants had received the FDC with dose session as (ambrisentan 10 milligram (mg) + tadalafil 40 mg): GSK3380154, TABA, Tablet Weight 560mg/2mg SLS, with reference to the 2 monotherapy components for ambrisentan 10 mg and tadalafil 40 mg, which were taken concurrently, which evaluated bioavailability. This was received as a single oral dose, under fasting condition and was followed by a wash-out period of 7-days, before the start of next dose F4.
- Part 1,Treatment F4: In the F4 arm of Part 1, the participants had received the FDC with dose session as (ambrisentan 10 milligram (mg) + tadalafil 40 mg): GSK3380154, TAB-A, Tablet Weight 560mg/4mg SLS, with reference to the 2 monotherapy components for ambrisentan 10 mg and tadalafil 40 mg, which were taken concurrently, which evaluated bioavailability. This was received as a single oral dose, under fasting condition and was followed by a wash-out period of 7-days, before the start of next dose R.
Arm/Group | Part 1,Treatment F1 | Part 1,Treatment F2 | Part 1,Treatment F3 | Part 1,Treatment F4 | Part 1, Treatment R
Number analyzed (Participants) | 21 | 23 | 23 | 22 | 21
Hour
  Ambrisentan, t1/2 | 16.74 (18.2) | 15.25 (19.2) | 15.76 (17.3) | 15.25 (20.0) | 16.08 (17.9)
  Tadalafil, t1/2 | 17.08 (30.4) | 17.76 (33.3) | 18.38 (33.3) | 18.48 (33.0) | 18.04 (30.4)

21. Secondary Outcome: Plasma t1/2 for Ambrisentan and Tadalafil in FDC and Reference Treatment Under Fed and Fasted Condition- Part 2
Description: t1/2 is defined as the time required by the concentration of the drug to reach half of its original value. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Groups:
- Part 2, Treatment R: Participants were administered 2 monotherapies ambrisentan and tadalafil concurrently. The tablets were taken as single oral dose, under fasting condition and was followed by a wash-out period of 7-days.
Arm/Group | Part 2, Treatment R | Part 2, Treatment FG1 | Part 2, Treatment FG2 | Part 2, Treatment FG3
Number analyzed (Participants) | 21 | 20 | 20 | 20
Hour
  Ambrisentan, t1/2 (n=21,20,20,20) | 15.19 (24.5) | 15.76 (33.3) | 15.39 (18.6) | 16.60 (34.4)
  Tadalafil, t1/2, (n=20,20,20,20): number analyzed (Participants) | 20 | 20 | 20 | 20
  Tadalafil, t1/2, (n=20,20,20,20) | 18.58 (30.6) | 18.63 (33.2) | 18.22 (33.2) | 17.98 (32.6)

22. Secondary Outcome: Plasma t1/2 for Ambrisentan and Tadalafil in FDC and Reference Treatment Under Fed and Fasted Condition- Part 3A
Description: t1/2 is defined as the time required by the concentration of the drug to reach half of its original value. The serial blood samples were assessed at specified timepoints.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 18, 24, 36, 48 and 72 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Part 3A,Treatment X1 | Part 3A,Treatment X2 | Part 3A,Treatment R1 | Part 3A,Treatment R2
Number analyzed (Participants) | 32 | 33 | 32 | 32
Hour
  Ambrisentan, t1/2 | 15.65 (16.7) | 15.42 (15.9) | 14.66 (13.7) | 15.63 (16.6)
  Tadalafil, t1/2 | 20.09 (34.4) | 19.85 (34.2) | 19.29 (33.4) | 19.86 (36.8)

23. Secondary Outcome: Plasma t1/2 for Ambrisentan and Tadalafil in FDC and Reference Treatment Under Fed and Fasted Condition- Part 3B
Description: as for outcome 22
Time Frame: Pre-dose, 0.5 hours, 1, 1.5, 2, 2.5, 4, 8, 12, 24, 36, 48, and 72 hours postdose
Population: PK parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Part 3B,Treatment Y1 | Part 3B,Treatment Y2 | Part 3B,Treatment R3 | Part 3B,Treatment R4
Number analyzed (Participants) | 30 | 31 | 31 | 30
Hour
  Ambrisentan, t1/2 | 16.39 (21.6) | 16.42 (17.1) | 16.15 (18.7) | 16.00 (19.7)
  Tadalafil, t1/2 | 20.27 (34.3) | 19.01 (31.1) | 20.34 (34.4) | 18.95 (30.8)

24. Secondary Outcome: Change From Baseline in Vital- Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP), Part 1
Description: Vital signs were measured in semi-supine position after 5 minutes rest and were assessed for SBP and DBP. Change from Baseline, was defined as value at post-Baseline visit minus the Baseline value. Baseline, was defined as Day 1. Safety population included all the participants enrolled into the study who received atleast one dose of investigational product.
Time Frame: Baseline and Up to Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliliters of Mercury
Arm/Group | Part 1,Treatment F1 | Part 1,Treatment F2 | Part 1,Treatment F3 | Part 1,Treatment F4 | Part 1, Treatment R
Number analyzed (Participants) | 21 | 23 | 23 | 22 | 21
Milliliters of Mercury
  DBP, 0.5 hour | -3.33 (6.626) | -3.54 (4.164) | -4.20 (5.622) | -2.86 (5.330) | -2.79 (7.737)
  DBP, 1 hour | -5.33 (6.516) | -4.72 (4.008) | -5.63 (3.938) | -5.73 (6.001) | -4.40 (4.705)
  DBP, 2 hour | -5.24 (7.118) | -5.28 (5.220) | -5.98 (3.632) | -7.27 (5.101) | -5.83 (4.856)
  DBP, 4 hour | -4.29 (5.205) | -5.72 (4.064) | -6.07 (6.031) | -7.09 (5.149) | -5.21 (6.059)
  DBP, 8 hour | -9.10 (9.963) | -6.67 (6.704) | -6.50 (5.610) | -9.68 (6.263) | -7.83 (6.487)
  DBP, 12 hour | -4.76 (7.604) | -6.16 (5.685) | -5.72 (5.994) | -8.18 (8.296) | -5.60 (7.687)
  DBP, 24 hour | -5.86 (7.004) | -4.50 (6.308) | -4.07 (5.792) | -5.59 (6.235) | -3.55 (5.987)
  DBP, 48 hour | -2.38 (5.232) | -1.02 (6.091) | -4.02 (6.589) | -4.18 (4.382) | -0.74 (6.644)
  DBP, 72 hour | 0.76 (5.845) | -0.67 (5.676) | 0.20 (7.371) | -1.73 (5.311) | -0.15 (6.556)
  SBP, 0.5 hour | -1.10 (7.521) | -3.22 (8.590) | -1.59 (5.441) | -3.68 (6.438) | -3.36 (4.953)
  SBP, 1 hour | -2.76 (8.153) | -4.13 (7.091) | -2.54 (7.662) | -6.00 (7.624) | -3.74 (6.549)
  SBP, 2 hour | -6.05 (9.822) | -5.39 (7.116) | -3.11 (6.098) | -6.91 (9.148) | -5.40 (4.543)
  SBP, 4 hour | -3.90 (7.143) | -7.30 (8.244) | -5.50 (5.671) | -6.59 (7.699) | -5.36 (7.892)
  SBP, 8 hour | -6.10 (8.770) | -5.48 (9.279) | -4.02 (7.346) | -10.55 (9.579) | -8.40 (8.434)
  SBP, 12 hour | 0.14 (8.755) | -0.84 (9.278) | 0.54 (9.720) | -4.77 (12.023) | -3.60 (8.185)
  SBP, 24 hour | -1.48 (6.541) | -3.17 (9.767) | 0.02 (7.770) | -3.82 (7.276) | -1.79 (6.758)
  SBP, 48 hour | 1.52 (9.052) | 2.39 (7.010) | 2.50 (8.577) | -0.64 (7.315) | -0.31 (8.710)
  SBP, 72 hour | 6.95 (7.048) | 3.52 (8.993) | 3.37 (8.801) | 4.18 (7.341) | 3.00 (7.854)

25. Secondary Outcome: Change From Baseline in Vital Signs-Heart Rate, Part 1
Description: Vital signs were measured in semi-supine position after 5 minutes rest and were assessed for Heart rate. Change from Baseline, was defined as value at post-Baseline visit minus the Baseline value. Baseline, was defined as Day 1.
Time Frame: Baseline and Up to Day 3
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1,Treatment F1 | Part 1,Treatment F2 | Part 1,Treatment F3 | Part 1,Treatment F4 | Part 1, Treatment R
Number analyzed (Participants) | 21 | 20 | 20 | 20 | 21
Beats per minute
  HR, 0.5 hour | 2.98 (4.766) | 2.89 (2.558) | 1.13 (3.181) | 2.98 (3.718) | 3.74 (4.024)
  HR, 1 hour | 3.79 (4.314) | 4.11 (2.620) | 2.48 (4.981) | 3.30 (3.112) | 4.17 (4.223)
  HR, 2 hour | 3.69 (5.451) | 4.41 (3.107) | 1.91 (4.562) | 2.48 (4.393) | 2.83 (4.127)
  HR, 4 hour | 3.26 (4.449) | 3.63 (3.331) | 1.52 (4.636) | 3.16 (5.176) | 2.12 (3.584)
  HR, 8 hour | 8.26 (6.488) | 7.93 (5.407) | 7.17 (6.583) | 6.11 (5.323) | 7.55 (5.522)
  HR, 12 hour | 10.40 (6.387) | 12.75 (6.141) | 10.48 (7.264) | 11.11 (7.687) | 10.83 (5.342)
  HR, 24 hour | 6.17 (4.498) | 7.02 (6.343) | 6.52 (5.371) | 5.61 (5.381) | 6.74 (7.915)
  HR, 48 hour | 9.21 (5.110) | 8.67 (6.539) | 7.57 (5.623) | 6.48 (5.302) | 7.69 (5.501)
  HR, 72 hour | 6.21 (4.665) | 7.54 (7.762) | 6.57 (7.789) | 5.57 (7.323) | 5.03 (6.014)

26. Secondary Outcome: Change From Baseline in Vital- Temperature, Part 1
Description: Vital signs were measured in semi-supine position after 5 minutes rest and were assessed for temperature. Change from Baseline, was defined as value at post-Baseline visit minus the Baseline value. Baseline, was defined as Day 1.
Time Frame: Baseline and Up to Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree celsius
Arm/Group | Part 1,Treatment F1 | Part 1,Treatment F2 | Part 1,Treatment F3 | Part 1,Treatment F4 | Part 1, Treatment R
Number analyzed (Participants) | 21 | 23 | 23 | 22 | 21
Degree celsius
  Temperature, 0.5 hour | -0.20 (0.220) | -0.05 (0.250) | -0.12 (0.233) | -0.18 (0.357) | -0.03 (0.201)
  Temperature, 1 hour | -0.15 (0.275) | -0.09 (0.343) | -0.07 (0.216) | -0.06 (0.426) | -0.12 (0.386)
  Temperature, 2 hour | -0.14 (0.271) | -0.16 (0.383) | -0.23 (0.392) | -0.04 (0.473) | -0.14 (0.393)
  Temperature, 4 hour | -0.28 (0.363) | -0.08 (0.326) | -0.17 (0.328) | -0.03 (0.331) | -0.10 (0.381)
  Temperature, 8 hour | -0.04 (0.460) | 0.03 (0.438) | -0.08 (0.400) | 0.08 (0.422) | 0.02 (0.408)
  Temperature, 12 hour | 0.09 (0.371) | 0.16 (0.386) | -0.03 (0.438) | 0.08 (0.405) | 0.02 (0.597)
  Temperature, 24 hour | -0.04 (0.273) | 0.03 (0.328) | 0.14 (0.390) | 0.13 (0.413) | 0.07 (0.543)
  Temperature, 48 hour | -0.01 (0.371) | 0.18 (0.404) | 0.01 (0.393) | 0.05 (0.571) | 0.16 (0.508)
  Temperature, 72 hour | 0.12 (0.351) | 0.03 (0.503) | -0.02 (0.392) | 0.10 (0.424) | 0.02 (0.506)

27. Secondary Outcome: Change From Baseline in Vital Signs-Respiratory Rate, Part 1
Description: Vital signs were measured in semi-supine position after 5 minutes rest and were assessed for Respiratory rate. Change from Baseline, was defined as value at post-Baseline visit minus the Baseline value. Baseline, was defined as Day 1.
Time Frame: Baseline and Up to Day 3
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 1,Treatment F1 | Part 1,Treatment F2 | Part 1,Treatment F3 | Part 1,Treatment F4 | Part 1, Treatment R
Number analyzed (Participants) | 21 | 20 | 20 | 20 | 21
Breaths per minute
  Respiratory rate, 0.5 hour | -0.5 (2.23) | -0.7 (2.38) | -0.1 (3.17) | 0.3 (1.88) | 1.1 (1.49)
  Respiratory rate, 1 hour | -0.5 (2.62) | -1.0 (2.69) | 0.0 (2.76) | 0.6 (2.72) | 0.6 (2.11)
  Respiratory rate, 2 hour | -0.0 (1.56) | -1.0 (2.08) | -0.2 (2.55) | 0.4 (2.48) | 0.5 (2.44)
  Respiratory rate, 4 hour | -1.0 (2.10) | -0.8 (1.98) | -0.5 (2.91) | 0.2 (2.54) | 0.4 (2.42)
  Respiratory rate, 8 hour | 0.1 (2.73) | 0.2 (2.33) | 0.0 (2.63) | 0.6 (2.42) | 0.6 (2.20)
  Respiratory rate, 12 hour | 0.5 (2.86) | 0.4 (1.81) | 0.3 (2.93) | 0.9 (2.94) | 1.7 (3.30)
  Respiratory rate, 24 hour | -0.5 (2.44) | -0.7 (2.22) | -0.4 (2.63) | -0.1 (2.35) | 1.0 (3.20)
  Respiratory rate, 48 hour | 0.2 (2.68) | -0.6 (2.52) | 0.4 (3.07) | -0.0 (2.55) | 0.3 (3.86)
  Respiratory rate, 72 hour | -0.8 (2.44) | -0.1 (3.38) | 0.7 (3.17) | 1.0 (2.60) | 0.8 (2.46)

28. Secondary Outcome: Change From Baseline in Vital- SBP and DBP, Part 2
Description: Vital signs were measured in semi-supine position after 5 minutes rest and were assessed for SBP and DBP. Change from Baseline, was defined as value at post-Baseline visit minus the Baseline value. Baseline, was defined as Day 1.
Time Frame: Baseline and Up to Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliliters of Mercury
Arm/Group | Part 2, Treatment R | Part 2, Treatment FG1 | Part 2, Treatment FG2 | Part 2, Treatment FG3
Number analyzed (Participants) | 21 | 20 | 20 | 20
Milliliters of Mercury
  DBP, 0.5 hour | -2.29 (5.396) | 0.28 (5.707) | -0.25 (5.564) | -1.00 (5.091)
  DBP, 1 hour | -4.71 (7.329) | -4.23 (5.686) | -4.55 (5.264) | -4.35 (5.703)
  DBP, 2 hour | -5.67 (7.073) | -4.98 (5.488) | -5.85 (5.974) | -7.05 (5.954)
  DBP, 4 hour | -4.10 (6.468) | -3.53 (7.159) | -3.90 (7.080) | -5.10 (6.131)
  DBP, 8 hour | -4.43 (8.603) | -2.58 (7.979) | -5.15 (6.917) | -5.65 (8.278)
  DBP, 12 hour | -3.76 (7.800) | -3.18 (5.669) | -2.25 (6.084) | -4.35 (5.912)
  DBP, 24 hour | -3.00 (7.342) | -1.03 (6.791) | -2.00 (6.318) | -5.25 (6.470)
  DBP, 48 hour | -3.29 (7.125) | 2.48 (6.451) | 1.35 (5.956) | 1.40 (4.901)
  DBP, 72 hour | 0.95 (8.399) | 3.23 (5.357) | 2.05 (6.671) | 1.50 (6.907)
  SBP, 0.5 hour | -1.57 (5.388) | 1.63 (5.314) | 2.90 (4.576) | -0.33 (4.913)
  SBP, 1 hour | -4.43 (8.996) | -3.93 (6.057) | -2.05 (8.000) | -1.98 (7.144)
  SBP, 2 hour | -5.52 (8.848) | -2.48 (5.683) | -1.45 (7.112) | -7.33 (9.574)
  SBP, 4 hour | -3.05 (7.561) | -2.13 (6.456) | -2.45 (7.082) | -5.58 (6.053)
  SBP, 8 hour | -5.43 (8.982) | -3.98 (7.046) | -2.35 (6.471) | -6.38 (8.617)
  SBP, 12 hour | -0.05 (7.292) | 4.38 (9.418) | 2.00 (6.951) | 0.83 (6.822)
  SBP, 24 hour | -2.95 (7.847) | -0.68 (8.307) | -0.30 (8.163) | -1.68 (6.218)
  SBP, 48 hour | -2.00 (5.820) | 4.78 (7.911) | 0.85 (8.570) | 2.08 (4.660)
  SBP, 72 hour | 4.14 (7.636) | 5.13 (7.609) | 5.00 (6.345) | 3.48 (8.367)

29. Secondary Outcome: Change From Baseline in Vital Signs-Heart Rate, Part 2
Description: Vital signs were measured in semi-supine position after 5 minutes rest and were assessed for Heart rate. Change from Baseline, was defined as value at post-Baseline visit minus the Baseline value. Baseline, was defined as Day 1. Safety population included all the participants enrolled into the study who received atleast one dose of investigational product.
Time Frame: Baseline and Up to Day 3
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2, Treatment R | Part 2, Treatment FG1 | Part 2, Treatment FG2 | Part 2, Treatment FG3
Number analyzed (Participants) | 21 | 20 | 20 | 20
Beats per minute
  HR, 0.5 hour | 1.45 (4.040) | 2.85 (4.934) | 1.95 (6.219) | 2.20 (3.975)
  HR, 1 hour | 3.12 (4.475) | 3.85 (4.665) | 5.10 (6.528) | 5.35 (3.208)
  HR, 2 hour | 3.21 (3.720) | 3.75 (6.568) | 2.75 (5.959) | 6.45 (6.039)
  HR, 4 hour | 3.36 (5.287) | 5.45 (11.978) | 3.20 (7.428) | 6.00 (5.978)
  HR, 8 hour | 9.36 (7.720) | 8.30 (7.596) | 6.55 (6.901) | 8.30 (9.234)
  HR, 12 hour | 17.21 (7.348) | 14.80 (9.512) | 15.50 (6.473) | 16.45 (6.669)
  HR, 24 hour | 6.74 (6.100) | 8.80 (6.031) | 8.00 (7.395) | 8.70 (7.388)
  HR, 48 hour | 6.79 (5.361) | 5.70 (4.697) | 5.10 (5.973) | 5.90 (4.599)
  HR, 72 hour | 9.40 (8.412) | 7.90 (8.534) | 7.80 (8.427) | 9.30 (7.153)

30. Secondary Outcome: Change From Baseline in Vital- Temperature, Part 2
Description: Vital signs were measured in semi-supine position after 5 minutes rest and were assessed for temperature. Change from Baseline, was defined as value at post-Baseline visit minus the Baseline value. Baseline, was defined as Day 1. Safety population included all the participants enrolled into the study who received atleast one dose of investigational product.
Time Frame: Baseline and Up to Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree celsius
Arm/Group | Part 2, Treatment R | Part 2, Treatment FG1 | Part 2, Treatment FG2 | Part 2, Treatment FG3
Number analyzed (Participants) | 21 | 20 | 20 | 20
Degree celsius
  Temperature, 0.5 hour | -0.07 (0.403) | -0.02 (0.281) | -0.05 (0.261) | -0.14 (0.339)
  Temperature, 1 hour | -0.13 (0.280) | -0.11 (0.301) | -0.01 (0.300) | -0.04 (0.342)
  Temperature, 2 hour | -0.12 (0.349) | -0.17 (0.279) | -0.03 (0.310) | -0.23 (0.397)
  Temperature, 4 hour | -0.01 (0.348) | -0.06 (0.366) | 0.03 (0.286) | -0.19 (0.399)
  Temperature, 8 hour | 0.02 (0.397) | -0.08 (0.375) | 0.05 (0.343) | 0.03 (0.425)
  Temperature, 12 hour | 0.20 (0.409) | 0.04 (0.437) | 0.09 (0.418) | 0.10 (0.494)
  Temperature, 24 hour | -0.06 (0.285) | -0.02 (0.373) | 0.24 (0.298) | 0.07 (0.400)
  Temperature, 48 hour | -0.06 (0.441) | -0.06 (0.312) | 0.03 (0.353) | -0.11 (0.488)
  Temperature, 72 hour | -0.09 (0.435) | -0.13 (0.490) | 0.05 (0.375) | 0.06 (0.366)

31. Secondary Outcome: Change From Baseline in Vital Signs-Respiratory Rate, Part 2
Description: as for outcome 27
Time Frame: Baseline and Up to Day 3
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 2, Treatment R | Part 2, Treatment FG1 | Part 2, Treatment FG2 | Part 2, Treatment FG3
Number analyzed (Participants) | 21 | 20 | 20 | 20
Breaths per minute
  Respiratory rate, 0.5 hour | 0.7 (2.92) | -0.7 (2.27) | 0.3 (2.85) | -1.1 (2.04)
  Respiratory rate, 1 hour | -0.9 (2.15) | -0.4 (2.56) | 0.3 (2.70) | -0.7 (2.21)
  Respiratory rate, 2 hour | -0.6 (3.32) | -1.2 (2.86) | 0.4 (3.41) | -1.1 (2.70)
  Respiratory rate, 4 hour | -0.1 (2.87) | -0.1 (3.34) | -0.1 (3.21) | -1.0 (2.50)
  Respiratory rate, 8 hour | 0.1 (3.00) | 0.5 (2.82) | 0.4 (2.37) | -0.5 (2.06)
  Respiratory rate, 12 hour | 0.8 (2.93) | 0.2 (2.46) | 0.8 (2.61) | -0.5 (2.87)
  Respiratory rate, 24 hour | -0.1 (3.00) | -0.3 (2.92) | 1.3 (2.70) | 0.4 (2.32)
  Respiratory rate, 48 hour | -0.5 (2.60) | -0.2 (2.14) | 0.7 (2.62) | -0.6 (2.24)
  Respiratory rate, 72 hour | 0.2 (2.79) | 0.6 (2.67) | 0.6 (2.91) | 0.6 (2.82)

32. Secondary Outcome: Change From Baseline in Vital- SBP and DBP, Part 3A
Description: Vital signs were measured in semi-supine position after 5 minutes rest and were assessed for SBP, DBP. Change from Baseline, was defined as value at post-Baseline visit minus the Baseline value. Baseline, was defined as Day 1.
Time Frame: Baseline and Up to Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliliters of Mercury
Arm/Group | Part 3A,Treatment X1 | Part 3A,Treatment X2 | Part 3A,Treatment R1 | Part 3A,Treatment R2
Number analyzed (Participants) | 32 | 33 | 32 | 32
Milliliters of Mercury
  DBP, 0.5 hour | -3.47 (6.724) | -0.36 (5.821) | -3.02 (7.779) | -1.45 (6.943)
  DBP, 1 hour | -6.69 (6.509) | -4.73 (6.418) | -5.86 (7.055) | -5.36 (7.768)
  DBP, 2 hour | -8.97 (7.104) | -6.03 (5.840) | -6.89 (6.173) | -6.05 (7.745)
  DBP, 4 hour | -8.75 (5.879) | -6.24 (6.148) | -10.30 (6.722) | -6.27 (7.799)
  DBP, 8 hour | -8.41 (7.088) | -7.76 (8.100) | -6.45 (8.865) | -8.20 (8.845)
  DBP, 12 hour | -7.25 (7.097) | -6.18 (8.080) | -7.67 (8.274) | -7.36 (9.886)
  DBP, 24 hour | -7.25 (7.033) | -4.27 (6.011) | -4.77 (7.168) | -5.89 (6.847)
  DBP, 48 hour | -2.41 (9.414) | -0.79 (7.730) | -1.89 (6.945) | -1.77 (7.503)
  DBP, 72 hour | -1.56 (6.361) | 1.24 (6.544) | -1.52 (9.187) | 0.80 (9.118)
  SBP, 0.5 hour | 5.75 (5.236) | -0.32 (8.074) | 4.55 (8.543) | 0.17 (5.822)
  SBP, 1 hour | 2.88 (7.478) | -4.14 (9.772) | 2.86 (9.186) | -1.95 (5.959)
  SBP, 2 hour | 0.28 (9.549) | -2.05 (8.873) | -0.08 (7.294) | -3.95 (6.990)
  SBP, 4 hour | -1.72 (7.699) | -4.35 (9.423) | -4.30 (8.270) | -4.77 (7.717)
  SBP, 8 hour | -5.06 (9.313) | -5.32 (10.608) | -5.23 (9.288) | -5.27 (7.975)
  SBP, 12 hour | -0.03 (8.372) | -0.47 (10.702) | -1.05 (9.116) | -1.58 (9.155)
  SBP, 24 hour | -0.78 (8.974) | -1.08 (10.400) | -2.48 (6.478) | -2.08 (7.106)
  SBP, 48 hour | 2.72 (8.437) | 1.68 (9.134) | 1.36 (7.927) | 0.80 (7.661)
  SBP, 72 hour | 1.81 (8.538) | 3.14 (11.277) | 3.86 (11.332) | 3.52 (6.752)

33. Secondary Outcome: Change From Baseline in Vital Signs-Heart Rate, Part 3A
Description: as for outcome 25
Time Frame: Baseline and Up to Day 3
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 3A,Treatment X1 | Part 3A,Treatment X2 | Part 3A,Treatment R1 | Part 3A,Treatment R2
Number analyzed (Participants) | 32 | 33 | 32 | 32
Beats per minute
  HR, 0.5 hour | 8.28 (5.785) | 2.64 (3.900) | 10.66 (4.717) | 2.81 (4.156)
  HR, 1 hour | 10.28 (6.108) | 5.52 (4.154) | 12.97 (6.573) | 4.66 (3.897)
  HR, 2 hour | 11.06 (5.891) | 4.61 (4.565) | 11.41 (6.439) | 4.16 (4.306)
  HR, 4 hour | 10.16 (6.491) | 5.06 (6.910) | 10.91 (5.431) | 4.44 (4.629)
  HR, 8 hour | 9.06 (5.872) | 10.79 (7.847) | 10.16 (7.407) | 8.56 (6.624)
  HR, 12 hour | 15.28 (10.232) | 15.91 (9.669) | 14.38 (10.204) | 16.38 (8.917)
  HR, 24 hour | 8.72 (5.341) | 8.73 (7.048) | 7.00 (6.673) | 7.28 (4.704)
  HR, 48 hour | 8.50 (4.465) | 9.45 (7.527) | 9.47 (7.301) | 8.03 (5.290)
  HR, 72 hour | 9.19 (6.708) | 10.91 (10.476) | 9.59 (9.088) | 10.03 (8.041)

34. Secondary Outcome: Change From Baseline in Vital- Temperature, Part 3A
Description: as for outcome 26
Time Frame: Baseline and Up to Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Part 3A,Treatment X1 | Part 3A,Treatment X2 | Part 3A,Treatment R1 | Part 3A,Treatment R2
Number analyzed (Participants) | 32 | 33 | 32 | 32
Degree Celsius
  Temperature, 0.5 hour | 0.21 (0.288) | 0.01 (0.344) | 0.15 (0.306) | 0.12 (0.303)
  Temperature, 1 hour | 0.18 (0.252) | 0.07 (0.315) | 0.12 (0.262) | 0.04 (0.282)
  Temperature, 2 hour | 0.26 (0.278) | 0.05 (0.268) | 0.10 (0.244) | 0.07 (0.317)
  Temperature, 4 hour | 0.18 (0.352) | 0.15 (0.299) | 0.16 (0.305) | -0.01 (0.402)
  Temperature, 8 hour | 0.21 (0.450) | 0.12 (0.425) | 0.15 (0.409) | 0.15 (0.504)
  Temperature, 12 hour | 0.22 (0.409) | 0.27 (0.392) | 0.09 (0.366) | 0.27 (0.492)
  Temperature, 24 hour | 0.29 (0.429) | 0.25 (0.351) | 0.06 (0.332) | 0.16 (0.362)
  Temperature, 48 hour | 0.34 (0.713) | 0.28 (0.473) | 0.12 (0.358) | 0.32 (0.327)
  Temperature, 72 hour | 0.18 (0.414) | 0.20 (0.334) | 0.10 (0.418) | 0.18 (0.520)

35. Secondary Outcome: Change From Baseline in Vital Signs-Respiratory Rate, Part 3A
Description: as for outcome 27
Time Frame: Baseline and Up to Day 3
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 3A,Treatment X1 | Part 3A,Treatment X2 | Part 3A,Treatment R1 | Part 3A,Treatment R2
Number analyzed (Participants) | 32 | 33 | 32 | 32
Breaths per minute
  Respiratory rate, 0.5 hour | 0.4 (2.51) | 0.8 (1.95) | 1.5 (2.66) | -0.2 (2.46)
  Respiratory rate, 1 hour | 0.9 (2.83) | 0.2 (2.57) | 0.8 (2.26) | -0.7 (2.13)
  Respiratory rate, 2 hour | 0.7 (2.72) | 0.7 (2.59) | 0.6 (2.30) | 0.2 (2.89)
  Respiratory rate, 4 hour | 0.6 (2.76) | 0.2 (2.21) | 1.1 (2.59) | 0.1 (2.31)
  Respiratory rate, 8 hour | 0.1 (2.85) | 0.1 (2.15) | 0.5 (2.49) | -0.3 (2.04)
  Respiratory rate, 12 hour | 0.9 (3.21) | 0.5 (2.33) | 0.6 (2.97) | 0.4 (3.11)
  Respiratory rate, 24 hour | -0.5 (3.14) | 0.1 (2.26) | 0.2 (2.75) | -1.3 (2.58)
  Respiratory rate, 48 hour | 0.0 (2.03) | -0.1 (2.45) | 0.6 (2.93) | -0.7 (2.07)
  Respiratory rate, 72 hour | 0.6 (2.79) | 0.3 (3.05) | 0.8 (1.96) | 0.1 (2.59)

36. Secondary Outcome: Change From Baseline in Vital- SBP and DBP, Part 3B
Description: as for outcome 28
Time Frame: Baseline and Up to Day 3
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliliters of Mercury
Arm/Group | Part 3B,Treatment Y1 | Part 3B,Treatment Y2 | Part 3B,Treatment R3 | Part 3B,Treatment R4
Number analyzed (Participants) | 30 | 31 | 32 | 30
Milliliters of Mercury
  DBP, 0.5 hour | -1.42 (6.365) | -2.15 (6.582) | -2.53 (5.507) | -1.53 (6.965)
  DBP, 1 hour | -3.92 (6.443) | -3.31 (5.569) | -3.41 (7.157) | -3.73 (6.027)
  DBP, 2 hour | -6.52 (10.758) | -5.92 (6.044) | -5.00 (5.651) | -5.70 (5.842)
  DBP, 4 hour | -5.02 (4.481) | -6.85 (5.455) | -6.56 (6.488) | -6.80 (6.884)
  DBP, 8 hour | -4.38 (8.616) | -6.56 (5.815) | -7.81 (6.258) | -7.23 (9.095)
  DBP, 12 hour | -3.38 (8.189) | -5.15 (6.431) | -5.88 (6.644) | -7.57 (6.494)
  DBP, 24 hour | -1.62 (6.464) | -4.05 (6.571) | -3.31 (5.118) | -4.90 (5.636)
  DBP, 48 hour | -0.65 (7.945) | -0.40 (6.512) | -0.41 (5.491) | -1.50 (7.405)
  DBP, 72 hour | 0.85 (7.594) | 0.31 (4.790) | -0.47 (6.074) | -0.93 (6.781)
  SBP, 0.5 hour | 0.77 (9.323) | -0.92 (8.734) | 0.30 (8.287) | 0.43 (5.157)
  SBP, 1 hour | -1.27 (8.463) | 0.11 (8.945) | -0.20 (7.893) | 0.17 (6.823)
  SBP, 2 hour | -0.57 (9.657) | -4.34 (10.254) | -1.98 (7.925) | -1.10 (4.845)
  SBP, 4 hour | -4.17 (8.680) | -3.92 (7.959) | -3.14 (5.501) | -5.60 (7.831)
  SBP, 8 hour | -2.87 (10.059) | -2.95 (11.644) | -3.05 (8.804) | -5.03 (7.294)
  SBP, 12 hour | 2.17 (11.075) | 0.11 (13.298) | 0.45 (7.846) | -1.03 (10.562)
  SBP, 24 hour | -0.13 (8.805) | -2.56 (8.996) | 0.36 (5.210) | -1.77 (8.458)
  SBP, 48 hour | 5.33 (8.963) | 0.50 (8.748) | 3.45 (6.139) | 1.87 (8.345)
  SBP, 72 hour | 2.80 (9.174) | 1.76 (8.922) | 2.76 (7.236) | 1.70 (9.502)

37. Secondary Outcome: Change From Baseline in Vital Signs-Heart Rate, Part 3B
Description: Vital signs were measured in semi-supine position after 5 minutes rest and were assessed for HR. Change from Baseline, was defined as value at post-Baseline visit minus the Baseline value. Baseline, was defined as Day 1.
Time Frame: Baseline and Up to Day 3
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 3B,Treatment Y1 | Part 3B,Treatment Y2 | Part 3B,Treatment R3 | Part 3B,Treatment R4
Number analyzed (Participants) | 30 | 31 | 32 | 30
Beats per minute
  HR, 0.5 hour | 3.05 (5.103) | 3.50 (4.911) | 2.61 (4.652) | 2.78 (4.928)
  HR, 1 hour | 6.05 (5.784) | 4.92 (5.496) | 5.70 (4.621) | 5.48 (7.515)
  HR, 2 hour | 6.08 (5.706) | 3.76 (5.524) | 5.67 (4.148) | 5.58 (7.157)
  HR, 4 hour | 4.85 (6.498) | 3.69 (7.253) | 4.95 (5.564) | 6.22 (4.836)
  HR, 8 hour | 9.65 (8.102) | 7.34 (6.462) | 7.23 (6.453) | 8.78 (8.137)
  HR, 12 hour | 15.85 (9.232) | 15.50 (6.925) | 13.89 (7.574) | 16.62 (7.800)
  HR, 24 hour | 8.02 (6.086) | 6.92 (6.162) | 7.77 (6.677) | 7.72 (5.700)
  HR, 48 hour | 9.72 (5.845) | 8.18 (6.657) | 8.08 (6.610) | 10.15 (9.207)
  HR, 72 hour | 10.78 (8.397) | 9.18 (7.853) | 7.37 (7.256) | 9.62 (7.245)

38. Secondary Outcome: Change From Baseline in Vital- Temperature, Part 3B
Description: as for outcome 26
Time Frame: Baseline and Up to Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Part 3B,Treatment Y1 | Part 3B,Treatment Y2 | Part 3B,Treatment R3 | Part 3B,Treatment R4
Number analyzed (Participants) | 30 | 31 | 32 | 30
Degree Celsius
  Temperature, 0.5 hour (n=30,31,32,30) | 0.06 (0.239) | 0.13 (0.329) | 0.11 (0.404) | 0.05 (0.256)
  Temperature, 1 hour (n=30,31,32,30) | 0.06 (0.275) | 0.07 (0.290) | 0.10 (0.330) | 0.09 (0.291)
  Temperature, 2 hour (n=29,31,32,30): number analyzed (Participants) | 29 | 31 | 32 | 30
  Temperature, 2 hour (n=29,31,32,30) | 0.05 (0.341) | 0.07 (0.330) | 0.09 (0.316) | 0.04 (0.233)
  Temperature, 4 hour(n=30,31,32,30) | 0.10 (0.371) | 0.05 (0.385) | 0.07 (0.430) | 0.09 (0.275)
  Temperature, 8 hour (n=30,31,32,30) | 0.29 (0.497) | 0.22 (0.419) | 0.23 (0.456) | 0.17 (0.502)
  Temperature, 12 hour (n=30,31,32,30) | 0.31 (0.470) | 0.39 (0.358) | 0.32 (0.463) | 0.45 (0.425)
  Temperature, 24 hour (n=30,31,32,30) | 0.34 (0.347) | 0.12 (0.453) | 0.23 (0.352) | 0.19 (0.420)
  Temperature, 48 hour (n=30,31,32,30) | 0.19 (0.448) | 0.13 (0.424) | 0.16 (0.456) | 0.22 (0.444)
  Temperature, 72 hour (n=30,31,31,30): number analyzed (Participants) | 30 | 31 | 31 | 30
  Temperature, 72 hour (n=30,31,31,30) | 0.33 (0.422) | 0.26 (0.446) | 0.14 (0.450) | 0.08 (0.377)

39. Secondary Outcome: Change From Baseline in Vital Signs-Respiratory Rate, Part 3-B
Description: as for outcome 27
Time Frame: Baseline and Up to Day 3
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 3B,Treatment Y1 | Part 3B,Treatment Y2 | Part 3B,Treatment R3 | Part 3B,Treatment R4
Number analyzed (Participants) | 30 | 31 | 32 | 30
Breaths per minute
  Respiratory rate, 0.5 hour (n=30,31,32,30) | -0.3 (2.78) | 0.4 (2.99) | -0.8 (3.08) | 0.8 (3.06)
  Respiratory rate, 1 hour (n=30,31,32,30) | -0.6 (2.88) | -0.7 (3.08) | -0.1 (2.98) | 0.2 (2.06)
  Respiratory rate, 2 hour (n=30,31,32,30) | -0.2 (2.93) | 0.6 (3.64) | -0.1 (3.20) | 0.6 (2.31)
  Respiratory rate, 4 hour (n=30,31,32,30) | 0.3 (2.68) | 0.1 (3.47) | -0.4 (2.85) | 0.5 (2.76)
  Respiratory rate, 8 hour(n=30,31,32,30) | 0.4 (2.50) | 0.9 (3.31) | 0.0 (3.41) | 0.5 (2.75)
  Respiratory rate, 12 hour (n=30,31,32,30) | -0.8 (2.67) | -0.3 (2.82) | 0.2 (2.96) | 1.1 (2.89)
  Respiratory rate, 24 hour(n=30,31,32,30) | -1.3 (3.29) | -0.7 (3.08) | -0.6 (2.50) | 0.1 (3.04)
  Respiratory rate, 48 hour(n=30,31,32,30) | -0.8 (2.81) | -0.0 (3.35) | -0.1 (3.15) | 1.2 (3.09)
  Respiratory rate, 72 hour (n=30,31,31,30): number analyzed (Participants) | 30 | 31 | 31 | 30
  Respiratory rate, 72 hour (n=30,31,31,30) | -0.1 (3.73) | -0.0 (2.95) | 0.2 (2.89) | 0.6 (2.85)

40. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings, -Part 1
Description: 12-lead ECG, was measured in semi-supine position after 5 minutes rest. The data for worst case post-baseline has been reported. Data values for the participants with abnormal clinically significant values are reported. Safety population was used for analysis.
Time Frame: Up to Day 3
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part 1,Treatment F1 | Part 1,Treatment F2 | Part 1,Treatment F3 | Part 1,Treatment F4 | Part 1, Treatment R
Number analyzed (Participants) | 21 | 23 | 23 | 22 | 21
Participants | 0 | 0 | 0 | 0 | 0

41. Secondary Outcome: Number of Participants With Abnormal ECG Findings, -Part 2
Description: 12-lead ECG, were measured in semi-supine position after 5 minutes rest. It was conducted as triplicate at screen and baseline, whereas single measure at other times, unless out of range then triplicates were performed. The data for worst case post-baseline has been reported. Data values for the participants with abnormal clinically significant values are reported. Safety population was used for analysis.
Time Frame: Up to Day 3
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part 2, Treatment R | Part 2, Treatment FG1 | Part 2, Treatment FG2 | Part 2, Treatment FG3
Number analyzed (Participants) | 21 | 20 | 20 | 20
Participants | 0 | 0 | 0 | 0

42. Secondary Outcome: Number of Participants With Abnormal ECG Findings, -Part 3A
Description: as for outcome 41
Time Frame: Up to Day 3
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part 3A,Treatment X1 | Part 3A,Treatment X2 | Part 3A,Treatment R1 | Part 3A,Treatment R2
Number analyzed (Participants) | 32 | 33 | 32 | 32
Participants | 0 | 0 | 0 | 0

43. Secondary Outcome: Number of Participants With Abnormal ECG Findings, -Part 3B
Description: as for outcome 41
Time Frame: Up to Day 3
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part 3B,Treatment Y1 | Part 3B,Treatment Y2 | Part 3B,Treatment R3 | Part 3B,Treatment R4
Number analyzed (Participants) | 30 | 31 | 32 | 30
Participants | 0 | 0 | 0 | 0

44. Secondary Outcome: Number of Participants With Hematology Values of Potential Clinical Importance (PCI)- Part1
Description: Blood samples were collected from the participants for analysis of hematology parameters like hematocrit, hemoglobin, lymphocytes, neutrophils, platelets and leukocytes. The data for number of participants, with low and high values of PCI have been reported. Safety population was used for analysis.
Time Frame: Up to Day 3
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 1,Treatment F1 | Part 1,Treatment F2 | Part 1,Treatment F3 | Part 1,Treatment F4 | Part 1, Treatment R
Number analyzed (Participants) | 21 | 23 | 23 | 22 | 21
Participants
  Hematocrit, low | 0 | 0 | 0 | 0 | 0
  Hematocrit, high | 0 | 0 | 0 | 0 | 0
  Hemoglobin, low | 0 | 0 | 0 | 0 | 0
  Hemoglobin, high | 0 | 0 | 0 | 0 | 1
  Lymphocytes, low | 0 | 1 | 0 | 0 | 0
  Lymphocyte, high | 0 | 0 | 0 | 0 | 0
  Neutrophils, low | 0 | 0 | 1 | 1 | 1
  Neutrophils, high | 0 | 0 | 0 | 0 | 0
  Platelets, low | 0 | 0 | 0 | 0 | 0
  Platelets, high | 0 | 0 | 0 | 0 | 0
  Leukocytes, low | 0 | 2 | 1 | 1 | 1
  Leukocytes, high | 0 | 0 | 0 | 0 | 0

45. Secondary Outcome: Number of Participants With Hematology Values of PCI - Part 2
Description: as for outcome 44
Time Frame: Day 2
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 2, Treatment R | Part 2, Treatment FG1 | Part 2, Treatment FG2 | Part 2, Treatment FG3
Number analyzed (Participants) | 21 | 20 | 20 | 20
Participants
  Hematocrit, low | 0 | 0 | 0 | 0
  Hematocrit, high | 0 | 0 | 0 | 0
  Hemoglobin, low | 0 | 0 | 0 | 0
  Hemoglobin, high | 0 | 0 | 0 | 0
  Lymphocytes, low | 0 | 0 | 0 | 0
  Lymphocytes, high | 0 | 0 | 0 | 0
  Neutrophils, low | 1 | 1 | 0 | 1
  Neutrophils, high | 0 | 0 | 0 | 0
  Platelets, low | 1 | 0 | 0 | 0
  Platelets, high | 0 | 0 | 0 | 00
  Leukocytes, low | 0 | 0 | 0 | 0
  Leukocytes, high | 0 | 0 | 0 | 0

46. Secondary Outcome: Number of Participants With Hematology Values of PCI - Part 3A
Description: Blood samples of 2 mL, via a cannula for were collected from the participants for analysis of hematology parameters like hematocrit, hemoglobin, lymphocytes, neutrophils, platelets and leukocytes. It was conducted at Day 2 (48 hours). The data for number of participants, with low and high values of PCI have been reported. Safety population was used for analysis.
Time Frame: Day 2
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 3A,Treatment X1 | Part 3A,Treatment X2 | Part 3A,Treatment R1 | Part 3A,Treatment R2
Number analyzed (Participants) | 32 | 33 | 32 | 32
Participants
  Hematocrit, low | 0 | 0 | 0 | 0
  Hematocrit, high | 0 | 0 | 0 | 0
  Hemoglobin, low | 0 | 0 | 0 | 0
  Hemoglobin, high | 0 | 0 | 0 | 0
  Lymphocytes, low | 1 | 1 | 0 | 0
  Lymphocytes, high | 0 | 0 | 0 | 0
  Neutrophils, low | 0 | 2 | 0 | 1
  Neutrophils, high | 0 | 0 | 0 | 0
  Platelets, low | 0 | 0 | 0 | 0
  Platelets, high | 0 | 0 | 0 | 0
  Leukocytes, low | 0 | 1 | 0 | 1
  Leukocytes, high | 0 | 0 | 0 | 0

47. Secondary Outcome: Number of Participants With Hematology Values of PCI - Part 3B
Description: Blood samples of 2 mL, via a cannula for were collected from the participants for analysis of hematology parameters like hematocrit, hemoglobin, lymphocytes, neutrophils, platelets and leukocytes. It was conducted at Day 2 (48 hour). The data for number of participants, with low and high values of PCI have been reported. Safety population was used for analysis.
Time Frame: Day 2
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 3B,Treatment Y1 | Part 3B,Treatment Y2 | Part 3B,Treatment R3 | Part 3B,Treatment R4
Number analyzed (Participants) | 30 | 31 | 32 | 30
Participants
  Hematocrit, low | 0 | 0 | 0 | 0
  Hematocrit, high | 0 | 0 | 0 | 0
  Hemoglobin, low | 0 | 0 | 0 | 0
  Hemoglobin, high | 0 | 0 | 0 | 0
  Lymphocytes, low | 0 | 0 | 0 | 0
  Lymphocytes, high | 0 | 0 | 0 | 0
  Neutrophils, low | 0 | 2 | 1 | 2
  Neutrophils, high | 0 | 0 | 0 | 0
  Platelets, low | 0 | 0 | 0 | 0
  Platelets, high | 0 | 0 | 0 | 0
  Leukocytes, low | 1 | 1 | 0 | 1
  Leukocytes, high | 0 | 0 | 0 | 0

48. Secondary Outcome: Number of Participants With Clinical Chemistry Values of PCI- Part1
Description: Blood samples of 2 mL, via a cannula for were collected from the participants for analysis of clinical chemistry parameters like glucose, calcium, albumin, sodium and potassium. The data for number of participants, with low and high values of PCI have been reported. Safety population was used for analysis.
Time Frame: Day 2
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part 1,Treatment F1 | Part 1,Treatment F2 | Part 1,Treatment F3 | Part 1,Treatment F4 | Part 1, Treatment R
Number analyzed (Participants) | 21 | 23 | 23 | 22 | 21
Participants
  Glucose, low | 0 | 0 | 0 | 0 | 0
  Glucose, high | 0 | 0 | 0 | 0 | 0
  Albumin, low | 0 | 0 | 0 | 0 | 0
  Albumin, high | 0 | 0 | 0 | 0 | 0
  Calcium, low | 0 | 0 | 0 | 0 | 0
  Calcium, high | 0 | 0 | 0 | 0 | 0
  Potassium, low | 0 | 0 | 0 | 0 | 0
  Potassium, high | 0 | 0 | 0 | 0 | 0
  Sodium, low | 0 | 0 | 0 | 0 | 0
  Sodium, high | 0 | 0 | 0 | 0 | 0

49. Secondary Outcome: Number of Participants With Clinical Chemistry Values of PCI- Part 2
Description: Blood samples of 2 mL, via a cannula for were collected from the participants for analysis of clinical chemistry parameters like glucose, calcium, albumin, sodium and potassium. It was collected at Day 2 (48 hour). The data for number of participants, with low and high values of PCI have been reported. Safety population was used for analysis.
Time Frame: Day 2
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 2, Treatment R | Part 2, Treatment FG1 | Part 2, Treatment FG2 | Part 2, Treatment FG3
Number analyzed (Participants) | 21 | 20 | 20 | 20
Participants
  Glucose, low | 0 | 0 | 0 | 0
  Glucose, high | 0 | 0 | 0 | 0
  Albumin, low | 0 | 0 | 0 | 0
  Albumin, high | 0 | 0 | 0 | 0
  Calcium, low | 0 | 0 | 0 | 0
  Calcium, high | 0 | 0 | 0 | 0
  Potassium, low | 0 | 0 | 0 | 0
  Potassium, high | 0 | 0 | 0 | 0
  Sodium, low | 0 | 0 | 0 | 0
  Sodium, high | 0 | 0 | 0 | 0

50. Secondary Outcome: Number of Participants With Clinical Chemistry Values of PCI- Part 3A
Description: Blood samples of 2 mL, via a cannula for were collected from the participants for analysis of clinical chemistry parameters like glucose, calcium, albumin, sodium and potassium. It was collected at (48 hour). The data for number of participants, with low and high values of PCI have been reported. Safety population was used for analysis.
Time Frame: Day 2
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 3A,Treatment X1 | Part 3A,Treatment X2 | Part 3A,Treatment R1 | Part 3A,Treatment R2
Number analyzed (Participants) | 32 | 33 | 32 | 32
Participants
  Glucose, low | 0 | 0 | 0 | 0
  Glucose, high | 0 | 0 | 0 | 0
  Albumin, low | 0 | 0 | 0 | 0
  Albumin, high | 0 | 0 | 0 | 0
  Calcium, low | 0 | 0 | 0 | 0
  Calcium, high | 0 | 0 | 0 | 0
  Potassium, low | 0 | 0 | 0 | 0
  Potassium, high | 0 | 0 | 0 | 0
  Sodium, low | 0 | 0 | 0 | 0
  Sodium, high | 0 | 0 | 0 | 0

51. Secondary Outcome: Number of Participants With Clinical Chemistry Values of PCI- Part 3B
Description: as for outcome 49
Time Frame: Day 2
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part 3B,Treatment Y1 | Part 3B,Treatment Y2 | Part 3B,Treatment R3 | Part 3B,Treatment R4
Number analyzed (Participants) | 30 | 31 | 32 | 30
Participants
  Glucose, low | 0 | 0 | 0 | 0
  Glucose, high | 0 | 0 | 0 | 0
  Albumin, low | 0 | 0 | 0 | 0
  Albumin, high | 0 | 0 | 0 | 0
  Calcium, low | 0 | 0 | 0 | 0
  Calcium, high | 0 | 0 | 0 | 0
  Potassium, low | 0 | 0 | 0 | 0
  Potassium, high | 1 | 0 | 0 | 0
  Sodium, low | 0 | 0 | 0 | 0
  Sodium, high | 0 | 0 | 0 | 0

52. Secondary Outcome: Number of Participants With Abnormal Urinalysis Results by Dipstick Method-Part 1
Description: Urine samples were collected at Day -1 (Baseline) and 48 hour, from the participants for urinalysis, by standard dipstick method. The parameters analyzed were ketones, glucose, occult blood, and protein. The number of participants with parameters detected as trace-lysed, trace-intact, trace, 2+ and 1+ was reported. Safety Population was used for analysis.
Time Frame: Up to Day 2
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 1,Treatment F1 | Part 1,Treatment F2 | Part 1,Treatment F3 | Part 1,Treatment F4 | Part 1, Treatment R
Number analyzed (Participants) | 21 | 23 | 23 | 22 | 21
Participants
  Ketone, trace-lysed, Day -1 | 0 | 0 | 0 | 0 | 0
  Ketone, trace-intact, Day -1 | 0 | 0 | 0 | 0 | 0
  Ketone, trace, Day -1 | 2 | 0 | 0 | 0 | 1
  Ketone, 2+, Day -1 | 0 | 0 | 0 | 0 | 0
  Ketone 1+, Day -1 | 0 | 0 | 0 | 0 | 0
  Ketone, trace-lysed, 48 hour | 0 | 0 | 0 | 0 | 0
  Ketone, trace-intact, 48 hour | 0 | 0 | 0 | 0 | 0
  Ketone, trace, 48 hour | 0 | 1 | 0 | 0 | 0
  Ketone, 2+, 48 hour | 0 | 0 | 0 | 0 | 0
  Ketone 1+, 48 hour | 0 | 0 | 0 | 0 | 0
  Glucose, trace-lysed, Day -1 | 0 | 0 | 0 | 0 | 0
  Glucose, trace-Intact, Day -1 | 0 | 0 | 0 | 0 | 0
  Glucose, trace, Day -1 | 0 | 0 | 0 | 0 | 0
  Glucose, 2+, Day -1 | 0 | 0 | 0 | 0 | 0
  Glucose, 1+, Day -1 | 0 | 0 | 0 | 0 | 0
  Glucose, trace-lysed, 48 hour | 0 | 0 | 0 | 0 | 0
  Glucose, trace-Intact, 48 hour | 0 | 0 | 0 | 0 | 0
  Glucose, trace, 48 hour | 0 | 0 | 0 | 0 | 0
  Glucose, 2+, 48 hour | 0 | 0 | 0 | 0 | 0
  Glucose, 1+, 48 hour | 0 | 0 | 0 | 0 | 0
  Occult blood, trace-lysed, Day -1 | 0 | 1 | 0 | 1 | 0
  Occult blood, trace-Intact, Day -1 | 0 | 1 | 0 | 1 | 1
  Occult blood, trace, Day -1 | 0 | 0 | 0 | 0 | 0
  Occult blood, 2+, Day -1 | 0 | 0 | 0 | 0 | 0
  Occult blood, 1+, Day -1 | 0 | 1 | 1 | 0 | 1
  Occult blood, trace-lysed, 48 hour | 1 | 1 | 0 | 1 | 0
  Occult blood, trace-Intact, 48 hour | 0 | 0 | 2 | 1 | 3
  Occult blood, trace, 48 hour | 0 | 0 | 0 | 0 | 0
  Occult blood, 2+, 48 hour | 0 | 0 | 0 | 0 | 0
  Occult blood, 1+, 48 hour | 2 | 1 | 0 | 0 | 0
  Protein, trace-lysed, Day -1 | 0 | 0 | 0 | 0 | 0
  Protein, trace-Intact, Day -1 | 0 | 0 | 0 | 0 | 0
  Protein, trace, Day -1 | 1 | 0 | 0 | 0 | 0
  Protein, 2+, Day -1 | 0 | 0 | 0 | 0 | 1
  Protein, 1+, Day -1 | 1 | 0 | 1 | 1 | 0
  Protein, trace-lysed, 48 hour | 0 | 0 | 0 | 0 | 0
  Protein, trace-Intact, 48 hour | 0 | 0 | 0 | 0 | 0
  Protein, trace, 48 hour | 0 | 0 | 0 | 0 | 1
  Protein, 2+, 48 hour | 0 | 0 | 0 | 0 | 0
  Protein, 1+, 48 hour | 0 | 0 | 0 | 0 | 0

53. Secondary Outcome: Number of Participants With Urinalysis Results by Dipstick Analysis-Part 2
Description: as for outcome 52
Time Frame: Up to Day 2
Population: Safety Population
Measure: Number; unit: Participants
Groups:
- Part 2, Treatment FG1: Participants were administered the FDC-G1 granulation size 1 (ambrisentan 10 milligram (mg) + tadalafil 40 mg) , from the formulation selected from Part 1. FG1 was administered as a single oral dose, under fasting condition and was followed by a wash-out period of 7-days, before the start of next dose FG2.
Arm/Group | Part 2, Treatment R | Part 2, Treatment FG1 | Part 2, Treatment FG2 | Part 2, Treatment FG3
Number analyzed (Participants) | 21 | 20 | 20 | 20
Participants
  Ketone, trace-intact, Day -1 | 0 | 0 | 0 | 0
  Ketone, trace, Day -1 | 1 | 2 | 2 | 1
  Ketone, 2+, Day -1 | 0 | 0 | 0 | 0
  Ketone, trace-intact, 48 hour | 0 | 0 | 0 | 0
  Ketone, trace, 48 hour | 1 | 0 | 1 | 0
  Ketone, 2+, 48 hour | 0 | 0 | 0 | 1
  Glucose, trace-Intact, Day -1 | 0 | 0 | 0 | 0
  Glucose, trace, Day -1 | 0 | 0 | 0 | 0
  Glucose, 2+, Day -1 | 0 | 0 | 0 | 0
  Glucose, trace-Intact, 48 hour | 0 | 0 | 0 | 0
  Glucose, trace, 48 hour | 0 | 0 | 0 | 0
  Glucose, 2+, 48 hour | 0 | 0 | 0 | 0
  Occult blood, trace-Intact, Day -1 | 0 | 1 | 0 | 1
  Occult blood, trace, Day -1 | 0 | 0 | 0 | 0
  Occult blood, 2+, Day -1 | 0 | 0 | 0 | 0
  Occult blood, trace-Intact, 48 hour | 0 | 0 | 0 | 1
  Occult blood, trace, 48 hour | 0 | 0 | 0 | 0
  Occult blood, 2+, 48 hour | 0 | 0 | 0 | 0
  Protein, trace-Intact, Day -1 | 0 | 0 | 0 | 0
  Protein, trace, Day -1 | 1 | 2 | 2 | 0
  Protein, 2+, Day -1 | 0 | 0 | 0 | 0
  Protein, trace-Intact, 48 hour | 0 | 0 | 0 | 0
  Protein, trace, 48 hour | 3 | 1 | 3 | 3
  Protein, 2+, 48 hour | 1 | 0 | 0 | 0

54. Secondary Outcome: Number of Participants With Urinalysis Results by Dipstick Analysis-Part 3A
Description: as for outcome 52
Time Frame: Up to Day 2
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part 3A,Treatment X1 | Part 3A,Treatment X2 | Part 3A,Treatment R1 | Part 3A,Treatment R2
Number analyzed (Participants) | 32 | 33 | 32 | 32
Participants
  Ketone, trace-lysed, Day -1 | 0 | 0 | 0 | 0
  Ketone, trace-intact, Day -1 | 0 | 0 | 0 | 0
  Ketone, trace, Day -1 | 4 | 3 | 4 | 4
  Ketone, 2+, Day -1 | 0 | 0 | 0 | 0
  Ketone 1+, Day -1 | 0 | 0 | 1 | 0
  Ketone, trace-lysed, 48 hour | 0 | 0 | 0 | 0
  Ketone, trace-intact, 48 hour | 0 | 0 | 0 | 0
  Ketone, trace, 48 hour | 2 | 1 | 1 | 3
  Ketone, 2+, 48 hour | 0 | 0 | 0 | 0
  Ketone 1+, 48 hour | 0 | 0 | 0 | 0
  Glucose, trace-lysed, Day -1 | 0 | 0 | 0 | 0
  Glucose, trace-Intact, Day -1 | 0 | 0 | 0 | 0
  Glucose, trace, Day -1 | 0 | 0 | 0 | 0
  Glucose, 2+, Day -1 | 0 | 0 | 0 | 0
  Glucose, 1+, Day -1 | 0 | 0 | 0 | 0
  Glucose, trace-lysed, 48 hour | 0 | 0 | 0 | 0
  Glucose, trace-Intact, 48 hour | 0 | 0 | 0 | 0
  Glucose, trace, 48 hour | 0 | 0 | 0 | 0
  Glucose, 2+, 48 hour | 0 | 0 | 0 | 0
  Glucose, 1+, 48 hour | 0 | 0 | 0 | 0
  Occult blood, trace-lysed, Day -1 | 3 | 6 | 4 | 3
  Occult blood, trace-Intact, Day -1 | 4 | 2 | 1 | 1
  Occult blood, trace, Day -1 | 0 | 0 | 0 | 0
  Occult blood, 2+, Day -1 | 0 | 1 | 2 | 0
  Occult blood, 1+, Day -1 | 0 | 0 | 0 | 0
  Occult blood, trace-lysed, 48 hour | 1 | 5 | 2 | 2
  Occult blood, trace-Intact, 48 hour | 3 | 0 | 1 | 0
  Occult blood, trace, 48 hour | 0 | 0 | 0 | 0
  Occult blood, 2+, 48 hour | 0 | 0 | 0 | 0
  Occult blood, 1+, 48 hour | 0 | 0 | 1 | 1
  Protein, trace-lysed, Day -1 | 0 | 0 | 0 | 0
  Protein, trace-Intact, Day -1 | 0 | 0 | 0 | 0
  Protein, trace, Day -1 | 1 | 0 | 0 | 2
  Protein, 2+, Day -1 | 0 | 0 | 0 | 0
  Protein, 1+, Day -1 | 0 | 0 | 0 | 0
  Protein, trace-lysed, 48 hour | 0 | 0 | 0 | 0
  Protein, trace-Intact, 48 hour | 0 | 0 | 0 | 0
  Protein, trace, 48 hour | 2 | 0 | 0 | 2
  Protein, 2+, 48 hour | 0 | 0 | 0 | 0
  Protein, 1+, 48 hour | 0 | 0 | 0 | 0

55. Secondary Outcome: Number of Participants With Urinalysis Results by Dipstick Analysis-Part 3B
Description: as for outcome 52
Time Frame: Up to Day 2
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 3B,Treatment Y1 | Part 3B,Treatment Y2 | Part 3B,Treatment R3 | Part 3B,Treatment R4
Number analyzed (Participants) | 30 | 31 | 32 | 30
Participants
  Ketone, trace-lysed, Day -1 | 0 | 0 | 0 | 0
  Ketone, trace-intact, Day -1 | 0 | 0 | 0 | 0
  Ketone, trace, Day -1 | 1 | 4 | 4 | 1
  Ketone, 3+, Day -1 | 0 | 1 | 0 | 0
  Ketone, trace-lysed, 48 hour | 0 | 0 | 0 | 0
  Ketone, trace-intact, 48 hour | 0 | 0 | 0 | 0
  Ketone, trace, 48 hour | 1 | 0 | 1 | 2
  Ketone, 3+, 48 hour | 0 | 0 | 0 | 0
  Glucose, trace-lysed, Day -1 | 0 | 0 | 0 | 0
  Glucose, trace-Intact, Day -1 | 0 | 0 | 0 | 0
  Glucose, trace, Day -1 | 0 | 0 | 0 | 0
  Glucose, 3+, Day -1 | 0 | 0 | 0 | 0
  Glucose, trace-lysed, 48 hour | 0 | 0 | 0 | 0
  Glucose, trace-Intact, 48 hour | 0 | 0 | 0 | 0
  Glucose, trace, 48 hour | 0 | 0 | 0 | 0
  Glucose, 3+, 48 hour | 0 | 0 | 0 | 0
  Occult blood, trace-lysed, Day -1 | 2 | 0 | 0 | 0
  Occult blood, trace-Intact, Day -1 | 0 | 1 | 3 | 1
  Occult blood, trace, Day -1 | 0 | 0 | 0 | 0
  Occult blood, 3+, Day -1 | 0 | 0 | 0 | 0
  Occult blood, trace-lysed, 48 hour | 0 | 0 | 0 | 0
  Occult blood, trace-Intact, 48 hour | 0 | 0 | 0 | 1
  Occult blood, trace, 48 hour | 0 | 0 | 0 | 0
  Occult blood, 3+, 48 hour | 1 | 0 | 0 | 0
  Protein, trace-lysed, Day -1 | 0 | 0 | 0 | 0
  Protein, trace-Intact, Day -1 | 0 | 0 | 0 | 0
  Protein, trace, Day -1 | 0 | 1 | 1 | 2
  Protein, 3+, Day -1 | 0 | 0 | 0 | 0
  Protein, trace-lysed, 48 hour | 0 | 0 | 0 | 0
  Protein, trace-Intact, 48 hour | 0 | 0 | 0 | 0
  Protein, trace, 48 hour | 2 | 1 | 0 | 1
  Protein, 3+, 48 hour | 0 | 0 | 0 | 0

56. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Adverse Events (AEs)-Part 1
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or is associated with liver injury and impaired liver function. Safety population was used for analysis.
Time Frame: Up to 42 days
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 1,Treatment F1 | Part 1,Treatment F2 | Part 1,Treatment F3 | Part 1,Treatment F4 | Part 1, Treatment R
Number analyzed (Participants) | 21 | 23 | 23 | 22 | 21
Participants
  Any SAE | 0 | 0 | 0 | 0 | 0
  Any AE | 12 | 13 | 13 | 15 | 12

57. Secondary Outcome: Number of Participants With SAEs and AEs-Part 2
Description: as for outcome 56
Time Frame: Up to 35 days
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part 2, Treatment R | Part 2, Treatment FG1 | Part 2, Treatment FG2 | Part 2, Treatment FG3
Number analyzed (Participants) | 21 | 20 | 20 | 20
Participants
  Any SAE | 0 | 0 | 0 | 0
  Any AE | 13 | 12 | 14 | 12

58. Secondary Outcome: Number of Participants With SAEs and AEs-Part 3A
Description: as for outcome 56
Time Frame: Up to 44 days
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part 3A,Treatment X1 | Part 3A,Treatment X2 | Part 3A,Treatment R1 | Part 3A,Treatment R2
Number analyzed (Participants) | 32 | 33 | 32 | 32
Participants
  Any SAE | 0 | 0 | 0 | 0
  Any AE | 24 | 21 | 25 | 23

59. Secondary Outcome: Number of Participants With SAEs and AEs-Part 3B
Description: as for outcome 56
Time Frame: Up to 44 days
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part 3B,Treatment Y1 | Part 3B,Treatment Y2 | Part 3B,Treatment R3 | Part 3B,Treatment R4
Number analyzed (Participants) | 30 | 31 | 32 | 30
Participants
  Any SAE | 0 | 0 | 0 | 0
  Any AE | 20 | 18 | 24 | 15

ADVERSE EVENTS:
Time Frame: All SAEs and AEs were collected from Day 1 to up to follow-up ( up to 165 days)
Description: Safety population included all the participants enrolled into the study who received atleast one dose of investigational product, was used to assess AE's and SAE's
Groups:
- Part 3A,Treatment X1: In the X1 arm of Part 3A, which evaluated the bioequivalence, the participants had received FDC (ambrisentan 10 mg + tadalafil 40 mg) either FG1, FG2 or FG3 (from granular formulation selected from Part 2), under fed state as a single oral dose. The fed state, particpants recived a high fat diet. This was followed by a wash-out period of 10-days, before the start of next dose X2.
Arm/Group | Part 1,Treatment F1 | Part 1,Treatment F2 | Part 1,Treatment F3 | Part 1,Treatment F4 | Part 1, Treatment R | Part 2, Treatment R | Part 2, Treatment FG1 | Part 2, Treatment FG2 | Part 2, Treatment FG3 | Part 3A,Treatment X1 | Part 3A,Treatment X2 | Part 3A,Treatment R1 | Part 3A,Treatment R2 | Part 3B,Treatment Y1 | Part 3B,Treatment Y2 | Part 3B,Treatment R3 | Part 3B,Treatment R4
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/23 | 0/23 | 0/22 | 0/21 | 0/21 | 0/20 | 0/20 | 0/20 | 0/32 | 0/33 | 0/32 | 0/32 | 0/30 | 0/31 | 0/32 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23 | 0/23 | 0/22 | 0/21 | 0/21 | 0/20 | 0/20 | 0/20 | 0/32 | 0/33 | 0/32 | 0/32 | 0/30 | 0/31 | 0/32 | 0/30
Other Adverse Events (participants affected / at risk) | 10/21 | 12/23 | 13/23 | 14/22 | 12/21 | 13/21 | 12/20 | 14/20 | 12/20 | 22/32 | 21/33 | 24/32 | 22/32 | 19/30 | 17/31 | 22/32 | 13/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1,Treatment F1 (N=21) | Part 1,Treatment F2 (N=23) | Part 1,Treatment F3 (N=23) | Part 1,Treatment F4 (N=22) | Part 1, Treatment R (N=21) | Part 2, Treatment R (N=21) | Part 2, Treatment FG1 (N=20) | Part 2, Treatment FG2 (N=20) | Part 2, Treatment FG3 (N=20) | Part 3A,Treatment X1 (N=32) | Part 3A,Treatment X2 (N=33) | Part 3A,Treatment R1 (N=32) | Part 3A,Treatment R2 (N=32) | Part 3B,Treatment Y1 (N=30) | Part 3B,Treatment Y2 (N=31) | Part 3B,Treatment R3 (N=32) | Part 3B,Treatment R4 (N=30)
Headache (Nervous system disorders) | 6 (6) | 11 (11) | 10 (10) | 13 (15) | 10 (12) | 13 (14) | 9 (10) | 13 (15) | 11 (11) | 17 (18) | 20 (21) | 22 (24) | 22 (23) | 18 (18) | 13 (13) | 16 (16) | 10 (10)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 5 (5) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 4 (4) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 5 (5) | 3 (3) | 2 (2) | 3 (3) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erection increased (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Priapism (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT02688387/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/87/NCT02688387/SAP_001.pdf